# Enhancing Recruitment, Linkage to Care and Treatment for HIV-Infected Men Who Have Sex with Men (MSM) in the United States

# A Study of the HIV Prevention Trials Network (HPTN)

# **Sponsored by:**

Division of AIDS (DAIDS)
United States (US) National Institute of Allergy and Infectious Diseases (NIAID)
US National Institute of Mental Health (NIMH)
US National Institute on Drug Abuse (NIDA)
US National Institutes of Health (NIH)

# **Protocol Chair:**

Chris Beyrer, MD, MPH Johns Hopkins University Baltimore, MD, USA

Protocol Co-Chair Robert H. Remien, PhD Columbia University New York, NY, USA

**DAIDS Document ID: 11995** 

Final Version 2.0 July 3, 2017

# **Enhancing Recruitment, Linkage to Care and Treatment for HIV-Infected Men Who Have Sex** with Men (MSM) in the United States

# **TABLE OF CONTENTS**

| LIST<br>PROT<br>INVE<br>SCHI | OF AB<br>FOCOL<br>STIGA<br>EMA | CONTENTSBREVIATIONS AND ACRONYMSTEAM ROSTERTOR SIGNATURE PAGETOF STUDY DESIGN | iv<br>v!<br>ix |
|---|---|---|---|
| 1.0 | INTR | ODUCTION | 1 |
| | 1.1<br>1.2 | Background and Prior Research Rationale | |
| 2.0 | STUL | DY OBJECTIVES AND DESIGN | 5 |
| | 2.1<br>2.2<br>2.3<br>2.4<br>2.5 | Primary Objectives Secondary Objectives Exploratory Objectives Modeling Objective Study Design | 5<br>6 |
| 3.0 | STUI | DY POPULATION | 7 |
| | 3.1<br>3.2<br>3.3<br>3.4<br>3.5<br>3.6<br>3.7 | Inclusion Criteria Exclusion Criteria Recruitment Process Co-Enrollment Guidelines Participant Retention Participant Withdrawal and Early Termination Study Sites | 8<br>8<br>8 |
| 4.0 | STUL | DY INTERVENTION | 10 |
| | 4.1<br>4.2<br>4.3 | Linkage to Care and ART Initiation (MyLife, MyChoices, MyCare (Step 1)). Adherence Counseling (MyCare (Step 2)) Communication, Retention and Follow-up (MyHealth) | 14 |
| 5.0 | STUL | DY PROCEDURES | 15 |
| | 5.1<br>5.2<br>5.3<br>5.4<br>5.5<br>5.6<br>5.7<br>5.8 | Screening Visits Enrollment Visit (M0) Tailored Communication Monthly Contact Follow-up Visits (M3, M6, M9, M12, M18) Final Visit (M24) Data Collection on ART Initiation and Visit Attendance Questionnaires | 16<br>16<br>16<br>17<br>17 |
| 6.0 | | TY MONITORING AND ADVERSE EVENT REPORTING | |
| | 6.1<br>6.2 | Safety Monitoring Social Impact Reporting | |

| 7.0 | STAT | TISTICAL CONSIDERATIONS | 20 |
|---|---|---|---|
| | 7.1 | Review of Study Design | 20 |
| | 7.2 | Endpoints | |
| | 7.3 | Accrual, Follow-up and Sample Size | |
| | 7.4 | Random Assignment | |
| | 7.5 | Blinding | |
| | 7.6 | Data Analysis | 23 |
| 8.0 | HUM | AN SUBJECTS CONSIDERATIONS | 26 |
| | 8.1 | Ethical Review | 26 |
| | 8.2 | Informed Consent | 26 |
| | 8.3 | Incentives | 26 |
| | 8.4 | Confidentiality | |
| | 8.5 | Communicable Disease Reporting Requirements | |
| | 8.6 | Study Discontinuation | 27 |
| 9.0 | LAB | ORATORY SPECIMENS AND BIOHARDS CONTAINMENT | 28 |
| | 9.1 | Local Laboratory Specimens | |
| | 9.2 | LC Specimens | |
| | 9.3 | Quality Control and Quality Assurance Procedures | |
| | 9.4 | QC for HIV Diagnostic Testing | |
| | 9.5 | Phylogenetic Analysis | |
| | 9.6 | Specimen Storage and Possible Future Research Testing | |
| | 9.7 | Biohazard Containment | |
| | 9.8 | Resistance Testing at Local Laboratories. | |
| 10.0 | | ELING COMPONENT | |
| | 10.1 | Background and Prior Research | |
| | 10.2 | Rationale | |
| | 10.3 | Model Population and Setting | |
| | 10.4 | Main Model Outcomes | |
| | 10.5 | Modeling Stages | |
| 11.0 | ADM | INISTRATIVE PROCEDURES | |
| | 11.1 | Protocol Registration | |
| | 11.2 | Study Activation | |
| | 11.3 | Study Coordination | |
| | 11.4 | Study Monitoring | |
| | 11.5 | Protocol Compliance | |
| | 11.6 | Investigator's Records | |
| | 11.7 | Use of Information and Publications | |
| 12.0 | | ERENCES | |
| | | Schedule of Study Visits, Evaluations and Procedures | |
| | | Schedule of Questionnaire Domain Administration | |
| Appe | ndix III | : Informed Consent Templates | 54 |
| Annei | ndix IV | : Tailored Case Management Intervention Components | 79 |

# Enhancing Recruitment, Linkage to Care and Treatment for HIV-Infected Men Who Have Sex with Men (MSM) in the United States

#### LIST OF ABBREVIATIONS AND ACRONYMS

ACA Affordable Care Act

AIDS Acquired Immunodeficiency Syndrome

ART antiretroviral therapy ARV antiretroviral drug

CAB Community Advisory Board

CCM Chronic Care Model

CD4 Cluster of Differentiation 4 (a glycoprotein found on the surface of T-helper cells that

serves as a receptor), in the context of this protocol, CD4+ refers to cells with this

glycoprotein)

CDC Centers for Disease Control and Prevention

CFR Code of Federal Regulations

CI confidence interval

CLIA Continuous Laboratory Improvement Act

CM Case Manager CRF case report form DAIDS Division of AIDS

DC-RDS deep-chain respondent driven sampling

DR direct recruitment EC Ethics Committee

FDA (United States) Food and Drug Administration

HCV Hepatitis C virus

HHS (United States Department of) Health and Human Services

HIV Human Immunodeficiency Virus HPTN HIV Prevention Trials Network

ID identification

ICF informed consent forms

ICH International Council for Harmonisation

IoR Investigator of Record
IRB Institutional Review Board
LC (HPTN) Laboratory Center

LDMS Laboratory Data Management System
LGBT Lesbian, gay, bisexual, and transgender
LOC (HPTN) Leadership and Operations Center
MMWR Morbidity and Mortality Weekly Report
MRC (HPTN) Manuscript Review Committee

MSM Men Who Have Sex with Men

NHBS National HIV Behavioral Surveillance

NIAID (United States) National Institute of Allergy and Infectious Diseases

NIDA (United States) National Institute on Drug Addiction

NIH (United States) National Institutes of Health

NSFG National Survey of Family Growth

NIMH (United States) National Institute of Mental Health

OHRP Office for Human Research Protections

PAF population attributable fraction PEP post-exposure prophylaxis

# **Enhancing Recruitment, Linkage to Care and Treatment for HIV-Infected Men Who Have Sex with Men (MSM) in the United States**

# LIST OF ABBREVIATIONS AND ACRONYMS (continued)

PF preventable fraction PrEP pre-exposure prophylaxis

PRO (DAIDS) Protocol Registration Office

PSRC (DAIDS) Prevention Science Review Committee PUMA Prevention Umbrella for MSM in the Americas

QA quality assurance QC quality control

RDS respondent driven sampling RSC Regulatory Support Center

SAMISS Substance Abuse/Mental Illness Symptoms Screener SDMC (HPTN) Statistical and Data Management Center

SES socio-economic status

SMC (HPTN) Study Monitoring Committee

SOC standard of care

SRC (HPTN) Scientific Review Committee

SSP Study Specific Procedures
STI Sexually Transmitted Infection
TasP Treatment as Prevention
UAI unprotected anal intercourse

US United States VL viral load

# Enhancing Recruitment, Linkage to Care and Treatment for HIV-Infected Men Who Have Sex with Men (MSM) in the United States

#### PROTOCOL TEAM ROSTER

#### Adeola Adeyeye, MD, MPA

Medical Officer

Prevention Science Program, DAIDS, NIAID,

NIH

Room 8B36 MSC 9832, 5601 Fishers Lane

Rockville, MD 20852 Phone: 240-669-5005

Email: adeyeyeao@niaid.nih.gov

#### Stefan Baral, MD, MPH, FRCPC

Associate Professor Department of Epidemiology Director, Key Populations Program Center for Public Health and Human Rights John Hopkins School of Public Health 615 N. Wolfe Street, Room E7146

Baltimore, MD 21205 Phone: 410-502-8975 Email: sbaral@jhsph.edu

#### Chris Beyrer, MD, MPH

Professor of Epidemiology, International Health, and Health, Behavior and Society Director, Center for Public Health and Human

Rights

Associate Director, Johns Hopkins Center for

**AIDS Research** 

Johns Hopkins University 615 N. Wolfe St, E 7152 Baltimore, MD, 21205

Phone: 410 614 5247 Email: <u>cbeyrer@jhu.edu</u>

### Marie-Claude Boily, PhD

Professor of Mathematical Epidemiology Department of Infectious Diseases Epidemiology School of Public Health Imperial College London Norfolk Place, St-Mary's Campus London, UK W2 1PG

Phone: 44-0-207-594-3263 Email: <u>mc.boily@ic.ac.uk</u>

#### Marcus D. Bolton, MEd

Sr. Community Programs Manager HPTN LOC, FHI 360 359 Blackwell St., Durham, NC 27701 Phone: 919-544-7040, Ex. 11678

Email: mbolton@fhi360.org

# Vanessa Cummings, B.S, MT (ASCP)

HPTN Laboratory Center QA/QC

Representative

Johns Hopkins Univ. School of Medicine

Pathology Building, Room 311

600 North Wolfe Street Baltimore, MD 21287

Phone: 410-614-0479

Email: vcummin1@jhmi.edu

#### Carlos Del Rio, MD

Emory Center for AIDS Research Ponce de Leon Center

341 Ponce de Leon Avenue, Northeast

Atlanta, GA 30308 Phone: 404-727-1557 Email: cdelrio@emory.edu

#### Dobromir Dimitrov, PhD

Senior Staff Scientist SCHARP-FHCRC 1100 Fairview Ave. N, M2-C200 PO Box 19024 Seattle, WA 98109

Phone: 206-667-1933 Email: dobromir@scharp.org

# Lynda Emel, PhD

Associate Director HPTN SDMC SCHARP-FHCRC 1100 Fairview Ave. N, E3-129 PO Box 19024 Seattle, WA 98109

Phone: 206-667-5803 Email: <u>lemel@scharp.org</u>

# Enhancing Recruitment, Linkage to Care and Treatment for HIV-Infected Men Who Have Sex with Men (MSM) in the United States

#### PROTOCOL TEAM ROSTER (Continued)

#### Susan Eshleman, MD, PhD

**HPTN Laboratory Center Virologist** Johns Hopkins Univ. School of Medicine 720 Rutland Ave. Ross Building, Room 646 Baltimore, MD, 21205

Phone: 410-614-4734 Email: seshlem@jhmi.edu

#### Jason Farley, PhD, MPH, ANP-BC, FAAN, **AACRN**

Associate Professor

Co-Director, Johns Hopkins Center for AIDS

Research

Department of Community-Public Health Johns Hopkins University School of Nursing 525 N. Wolfe Street

Baltimore, MD 21205 Phone: 410-502-7563 Email: <u>ifarley1@jhu.edu</u>

#### Theresa Gamble, PhD

Scientist II

HPTN LOC, FHI 360

359 Blackwell St. Durham, NC 27701 Phone: 919-544-7040, Ex. 11350 Email: tgamble@fhi360.org

#### James Hughes, PhD

Professor of Biostatistics University of Washington Mailstop 357232

Seattle, WA 98195 Phone: 206-616-2721

Email: jphughes@u.washington.edu

#### Risha Irvin, MD, MPH

**Assistant Professor** 

Division of Infectious Diseases Johns Hopkins University

Fisher Center for Environmental Infectious

Diseases

725 N Wolfe Street, Room 218A

Baltimore, MD 21205 Phone: 443-287-4843 Email: rirvin1@jhmi.edu

#### Anna LeViere, MPH

Clinical Research Manager HPTN LOC, FHI 360 359 Blackwell St. Durham, NC 27701

Phone: 919-544-7040, Ex. 11585

Email: aleviere@fhi360.org

#### Kenneth Mayer, MD

Infectious Disease Attending and Director of HIV

Prevention Research

Beth Israel Deaconess Medical Center

Professor of Medicine Harvard Medical School Medical Research Director

The Fenway Institute, Fenway Health

Boston, MA 02215 Phone: 617-927-6087

Email: Khmayer@gmail.com

# Laura A. McKinstry, MPH

Clinical Data Manager

Statistical Center for HIV/AIDS Research and

Prevention (SCHARP)

Vaccine and Infectious Disease Division (VIDD)

1100 Fairview Avenue North E3-129

PO Box 19024 Seattle, WA 98109 Phone: 206.667.7322

Email: lamckins@scharp.org

# **Enhancing Recruitment, Linkage to Care and Treatment for HIV-Infected Men Who Have Sex with Men (MSM) in the United States**

#### PROTOCOL TEAM ROSTER (Continued)

#### Greg Millett, MPH

Vice President and Director, Public Policy amfAR 1150 17th Street, NW Suite 406

Washington, DC 20036 Phone: 202-331-8600

Email: Greg.Millett@amfar.org

#### Kate Mitchell, PhD

Research Fellow Imperial College London Department of Infectious Diseases Epidemiology School of Public Health Imperial College London Norfolk Place, St-Mary's Campus London, UK W2 1PG

Email: kate.mitchell@imperial.ac.uk

#### E. Turner Overton, MD

University of Alabama at Birmingham 1530 3rd Ave S CCB Rm 330A Birmingham, AL 35294 Phone: 205-966-2373

Email: toverton@uab.edu

#### Robert H. Remien, PhD

Professor of Clinical Psychology (in Psychiatry)
Director, HIV Center for Clinical and
Behavioral Studies
Associate Director, Division of Gender,
Sexuality and Health, NY State Psychiatric
Institute and Columbia University
722 West 168th Street, Floor R3, Room 308
New York, NY 10032

Phone: 646-774-6933

Email: <u>rhr1@cumc.columbia.edu</u>

#### Paul Richardson, MSc

Senior QA/QC Coordinator HPTN LC Johns Hopkins Univ. Dept. of Pathology Pathology Building, Room 306 600 North Wolfe Street Baltimore, MD 21287 Phone: 410-502-0435 Email: pricha18@jhmi.edu

# Ethan Wilson

Statistical Research Associate Statistical Center for HIV/AIDS Research and Prevention (SCHARP) Fred Hutchinson Cancer Research Center 1100 Fairview Ave. N., Mail Stop M2-C200 Seattle, WA 98109

Phone: 206.667.7207 Email: eawilson@fredhutch.org

#### Patrick Wilson, PhD

Associate Professor of Sociomedical Sciences Columbia University Mailman School of Public Health 722 W. 168th Street, 5th Floor New York, NY 10032 Phone: 212-305-1852

Email: pw2219@columbia.edu

# Enhancing Recruitment, Linkage to Care and Treatment for HIV-Infected Men Who Have Sex with Men (MSM) in the United States

#### Version 2.0 / July 3, 2017 INVESTIGATOR SIGNATURE PAGE

A Study of the HIV Prevention Trials Network (HPTN)

#### Sponsored by:

Division of AIDS (DAIDS)
United States (US) National Institute of Allergy and Infectious Diseases (NIAID)
US National Institute of Mental Health (NIMH)
US National Institute on Drug Abuse (NIDA)
US National Institutes of Health (NIH)

I, the Investigator of Record (IoR), agree to conduct this study in full accordance with the provisions of this protocol, including all appendices, as well as in compliance with United States (US) Health and Human Service regulations (45 Code of Federal Regulations [CFR] 46); applicable US Food and Drug Administration (FDA) regulations; standards of the International Conference on Harmonisation (ICH) Good Clinical Practices (E6); Institutional Review Board (IRB)/Ethics Committee (EC) determinations; all applicable in-country, state and local laws and regulations; and other applicable requirements (e.g., US National Institutes of Health, Division of AIDS) and institutional policies. I agree to maintain all study documentation for a minimum of three years after submission of the site's final Financial Status Report to the Division of AIDS (DAIDS), unless otherwise specified by DAIDS or the HIV Prevention Trials Network (HPTN) Leadership and Operations Center (LOC). Publication of the results of this study will be governed by HPTN policies. Any presentation, abstract, or manuscript will be submitted to the HPTN Manuscript Review Committee (MRC) and the Division of AIDS (DAIDS) for review prior to submission.

I have read and understand the information in this protocol and will ensure that all associates, colleagues, and employees assisting in the conduct of the study are informed about the obligations incurred by their contribution to the study.

| Name of Site Investigator of Record | |
|------------------------------------------|------|
| Signature of Site Investigator of Record | Date |

# Enhancing Recruitment, Linkage to Care and Treatment for HIV-Infected Men Who Have Sex with Men (MSM) in the United States

#### **SCHEMA**

**Purpose:** 

The purpose of this study is to develop and assess the efficacy of an integrated strategy that includes feasible and scalable interventions to identify, recruit, link to care, retain in care, attain, and maintain viral suppression among HIV-infected men who have sex with men (MSM) in the United States (US).

Design:

This study will use deep-chain respondent driven sampling (DC-RDS) and direct recruitment (DR) to identify and recruit HIV-infected MSM who are not virally suppressed. A subset of these men will be enrolled into one of two study arms. The intervention arm will provide a Case Manager (CM) intervention package designed to enhance linkage to care, antiretroviral treatment (ART) initiation, treatment adherence and retention in care. The control arm will provide the standard of care (SOC) for linkage to care, initiation of ART, treatment adherence and retention in care. The primary outcome of the study is viral suppression, 24 months after enrollment. Phylogenetic methods will be used to evaluate the relationship between viruses in study participants. Mathematical modeling will be performed using demographic, behavioral, and clinical data generated from this study and other sources to estimate the population-level impact of the CM intervention on HIV incidence and to estimate the level of identification, linkage, ART coverage and viral suppression that would be required to achieve a substantial reduction in HIV incidence among MSM in the US settings where the study is conducted.

**Intervention:** 

The study intervention [MyLife, MyChoices, MyCare (Step 1), MyCare (Step 2), and MyHealth] is a program designed to enhance linkage, ART initiation, adherence and retention in care for MSM diagnosed with HIV. It will be administered by a trained CM and will include health care and supportive services navigation, adherence counseling, and tailored support for care engagement and treatment adherence.

**Population:** 

HIV-infected and HIV-uninfected adolescent (> 16 years old) and adult MSM, including transgender women, in selected US cities will be screened for this study. Enrollment will be limited to HIV-infected men who are not virally suppressed.

**Study Size:** 

Approximately 2700 MSM will be identified and recruited using a DC-RDS and DR strategies in four cities; 356 HIV-infected MSM who are not virally suppressed will be randomized (1:1) to the CM intervention and SOC control study arms of the study.

**Study Regimen:** There are no specific drug regimens under investigation in this study.

Study Duration: The overall study duration is 60 months: 24 months for DC-RDS recruitment and enrollment; 24 months of follow-up for participants who are randomized into the CM intervention and SOC control study arms; and approximately 12 months after the completion of participant study visits for data analyses, phylogenetic assessments and modeling.

**Study Sites:** 

Alabama Vaccine Research Center (Birmingham, AL); Fenway Health (Boston, MA); Johns Hopkins Adult AIDS (Baltimore, MD); and the Ponce de Leon Ctr (Atlanta, GA)

# **Enhancing Recruitment, Linkage to Care and Treatment for HIV-Infected Men Who Have Sex with Men (MSM) in the United States**

#### **SCHEMA (Continued)**

# **Primary Objectives:**

- Assess the ability of DC-RDS to identify and recruit HIV-infected MSM in the US who are not virally suppressed.
- Compare the efficacy of the two study arms (CM intervention vs. SOC control) in achieving durable viral suppression (defined as HIV VL < 200 copies/ml) 24 months after enrollment.

#### **Secondary Objectives:**

- Assess HIV prevalence and the proportion of HIV-infected men who are virally suppressed by comparing early wave (approximately 1-6) vs. later (deep) wave (approximately 7-12) DC-RDS participants.
- Compare the proportion of men in the two study arms who are virally suppressed at 3, 6, 9, 12 and 18 months after enrollment.
- Assess linkage to care and retention in care in the two study arms by comparing the 1) proportion of men with at least one care visit within 30 days of enrollment, 2) time to the first care visit, and 3) proportion of men with at least four care visits (one in each six-month interval, with at least 60 days between these visits) over the 24 months after enrollment.
- Compare the proportion of men with HIV-hepatitis C virus (HCV) co-infection in the two study arms who are linked to care (defined as one care visit within 30 days of enrollment) and who achieve (HIV) viral suppression 24 months after enrollment.
- Examine the association between baseline behavioral, socio-demographic, and clinical characteristics (including syphilis) of HIV-infected men and viral suppression status for all men screened via DC-RDS and for the men in the two study arms 24 months after enrollment.
- Compare the two study arms with respect to ART adherence at 24 months after enrollment and changes in sexual risk behavior, health care utilization, stigma, substance use and mental health from baseline to 24 months after enrollment.
- Evaluate the feasibility and scalability of the CM intervention by measuring the number of intervention contacts (e.g., text message, email, phone, in person) per participant over 24 months.
- Compare the experience of linkage to and ongoing HIV care among participants in the two study arms by conducting and analyzing exit interviews with participants and CMs.

# **Enhancing Recruitment, Linkage to Care and Treatment for HIV-Infected Men Who Have Sex with Men (MSM) in the United States**

#### **SCHEMA (Continued)**

# **Exploratory Objectives:**

- Use phylogenetic methods to evaluate the relationship between HIV strains in study participants. Men who were likely to have been recently infected at enrollment will be identified using a multi-assay algorithm. Evaluate the relationship of behavioral, sociodemographic, and clinical characteristics to viral networks (e.g., clusters, linked infections).
- Use laboratory assessments to characterize the study cohort and to evaluate the impacts of study interventions. These assessments may include analysis of HIV drug resistance and antiretroviral (ARV) drug use. Additional analyses may be conducted to analyze HCV strains, including phylogenetic analysis of HCV. Samples from this study may also be used to evaluate the performance of assays related to HIV and HCV infection.

# **Modeling Objective:**

• Develop, calibrate, and use a mathematical model of HIV transmission among MSM in the US to assess the short and long-term population-level impact of the study strategy, and its independent CM intervention components (e.g., HIV testing, ART uptake, retention in care and viral suppression), on HIV incidence and to estimate the level of viral suppression required to reduce HIV incidence in the MSM community by 10%, 20%, 30%, and 50% over 2, 5 and 10 years, and the likelihood of and time to elimination.

# Enhancing Recruitment, Linkage to Care and Treatment for HIV-Infected Men Who Have Sex with Men (MSM) in the United States OVERVIEW OF STUDY DESIGN



DC-RDS: Deep-Chain Respondent Driven Sampling DR: Direct Recruitment

HPTN 078, Final Version 2.0

July 3, 2017

#### 1.0 INTRODUCTION

#### 1.1 Background and Prior Research

The United States (US) is currently undergoing a widespread and severe HIV epidemic among gay, bisexual, and other men who have sex with men (MSM), which has been underway since at least 2003. In their most recent report, the US Centers for Disease Control and Prevention (CDC) reported that 62% of all new infections in the US were among MSM, a group who represent at most 2-4% of US adult men, and 1-2% of all adults. The US epidemic is strikingly concentrated in MSM populations—the only group among whom HIV infections burdens were rising in 2011. This epidemic is characterized by marked racial and ethnic disparities, with the highest HIV burdens among Black MSM, followed by Latino MSM.<sup>3</sup> The US MSM epidemic is marked by much higher incidence densities among the youngest MSM, those aged 13-24.4 HPTN 061, an incidence study in Black MSM, found a 3% incidence rate overall in this population, with a 5.9% incidence rate in those 18 to 29 years old. There is also a marked geographic component to the US epidemic among MSM, with the highest rates of incident HIV infection in Black, Latino, and White MSM found in the South. These health disparities are not limited to HIV prevalence and incidence burdens, but rather are also seen in lower rates of regular HIV testing, in lack of awareness of HIV status, in late presentation for HIV care, in poor adherence to antiretroviral therapy (ART), and in the failure to achieve viral suppression.<sup>3</sup>

The continuum of care, or cascade of care, has been useful to help characterize HIV burdens and understand gaps in HIV responses. The CDC estimate for the US population as a whole is that of the 1.2 million estimated persons living with HIV infection, 1 in 7 do not know they are living with HIV, only 4 in 10 are in care, and only 3 in 10 have sustained viral suppression.<sup>6</sup> African American MSM do less well across each step of this continuum, with an overall outcome of being half as likely to be fully virally suppressed if living with HIV infection compared to men of all other racial/ethnic categories.3 To address these health disparities, and to improve responses for gay and other MSM it is critical to reach higher proportions of HIV-infected MSM who are not virally suppressed, enhance their linkage to care, and increase the proportion of these men who can achieve, and maintain, HIV suppression. Intervention strategies and packages that can achieve these goals must be acceptable, feasible and scalable. This study will attempt to address two critical steps in the continuum of care for MSM in the US: enhanced outreach and recruitment of MSM living with HIV infection but not virally suppressed through deep-chain respondent driven sampling (DC-RDS); and enhanced treatment and care to increase the proportion of MSM who achieve sustained viral suppression through a case management (CM) intervention.

#### 1.1.1 The Need to Enhance Recruitment

The US CDC estimates that 14% of Americans living with HIV infection remain undiagnosed and unaware of their HIV infection status.<sup>6</sup> An additional 60% of those living with HIV are not currently in HIV care<sup>6</sup>—meaning that almost 70% of persons in the US with HIV infection are not currently on treatment or virally suppressed. This is a challenge for the health of these individuals, but also represents a pool of untreated HIV infections that drive ongoing transmission. Despite active testing and outreach campaigns in many jurisdictions, uptake of HIV testing remains too low in many communities, including among MSM, and is particularly challenging in minority communities and among younger age groups of MSM. Black MSM are nearly 5 fold less likely to have had a recent HIV test compared to White MSM in the US.<sup>3</sup> Active recruitment, and the use of innovative techniques for recruitment, is an urgent HIV research priority for controlling HIV infection among MSM.


Respondent driven sampling (RDS) has demonstrated effectiveness in reaching hard to sample populations, including among minority and low socio-economic status (SES) MSM in the US. Long Chain RDS, where referral chains are maintained over long waves of recruitment, is an innovative approach that has the potential to reach more hidden, marginalized and HIV-untested, unlinked, and not virally suppressed MSM living with HIV infection.

# 1.1.2 Deep-Chain Respondent Driven Sampling (DC-RDS)

RDS relies on the identification and enumeration of a discrete number of "seeds" who are incentivized to refer members of their social or sexual networks, who then repeat the process, generating successive waves of recruitment. RDS has been used successfully in the US and abroad to recruit marginalized MSM. RDS studies have reported success in recruiting MSM who have very low incomes, are homeless, men engaged in sex work, non-gay-identified and/or bisexually active men.<sup>7,8</sup> Moreover, studies that have used RDS to recruit black MSM in the US consistently find substantial proportions of HIV infected but untreated MSM in each respective study.<sup>8-10</sup> These studies obtained fairly similar samples despite varying demographics and risk profiles among initial seeds across the studies. This suggests that RDS can be a useful recruitment tool for research on marginalized populations and a method that has demonstrated considerable success in doing so in the US context, which is the focus of the proposed HPTN 078 study.

DC-RDS, also referred to as long chain RDS, where recruitment chains continue to propagate beyond the standard sixth wave of recruitment, has shown the potential to reach the most marginalized subsets of study participants, hence our interest in using this approach as a recruitment tool. <sup>11, 12</sup> A novel secondary aim of the study will be to compare early (approximately wave 1-6) versus later (approximately wave 7-12) recruitment waves to assess the ability of DC-RDS to identify HIV-infected MSM who are not virally suppressed in the selected cities.

#### 1.1.3 Evidence for Effectiveness of Early ART

There is strong biological plausibility that effective early ART can reduce sexual transmission of HIV between MSM by decreasing HIV viral load and, hence, infectiousness. Ecological evidence from San Francisco suggests that early ART initiation and high levels of treatment coverage may be associated with decreases in new HIV infections among MSM at population levels. <sup>13</sup> However, the ecological and other epidemiologic data are mixed, and recent reports from the United Kingdom and from France suggest rising rates of HIV infection in MSM despite high ART coverage of HIV-infected men in care. <sup>14, 15</sup>

In HPTN 052<sup>16</sup>, early ART initiation was confirmed to have high efficacy in preventing transmission among HIV serodiscordant couples. However, only 37 male-male discordant couples were recruited into HPTN 052 – with only one male-male couple in the US. Furthermore, recent epidemiologic and modeling data suggest that, in many populations of MSM, primary partnerships account for only a minority (30-35% in the PUMA [Prevention Umbrella for MSM in the Americas] modeling estimates) of HIV transmissions, with the majority occurring between non-primary sexual partners.<sup>17</sup> Thus, the population-level effectiveness of ART as HIV prevention among MSM is unknown and may not be measured most effectively through approaches based on discordant couples. Enhanced treatment of HIV-infected men within networks and at community levels may be important in reducing the spread of the epidemic among MSM.

# 1.1.4 Engagement in Care among MSM in the US

As there is a dearth of research on engagement-in-care strategies specific to the MSM population, challenges remain particularly prevalent among minority MSM in the US. Health care system navigation may offer a promising engagement-in-care strategy for MSM. Among young MSM of color there is a particular need for strengthened and tailored strategies for retention in care with links to social supportive services due to the multiple challenges in this group (e.g., access to health care, poverty, unemployment, stigma). 19-21

# 1.1.5 Interventions to Optimize Retention and Adherence

It is established that a combination of components and strategies best addresses challenges to HIV treatment and care; thus, the intervention package for linkage, retention and treatment adherence, with case management at its core, will draw from several evidence-based interventions. <sup>22-25</sup> The Care Coordination Model as outlined by Craig et al in 2011<sup>26</sup> has been shown to optimize linkage to and retention in care. <sup>27-29</sup> With the advent of the Affordable Care Act (ACA), and the uncertainty about the continuation of the ACA in some states, care coordination must include negotiating affordable care options available to study participants.

Behavioral interventions with the strongest beneficial impact on treatment adherence are cognitive-behavioral counseling interventions with a primary focus on treatment adherence.<sup>30-32</sup> In these sessions, patients are provided with <u>tailored</u> counseling to focus on problem solving and communication to address risk reduction, HIV disclosure, social support for adherence, and barriers to ART adherence.<sup>32-34</sup>

Use of mobile technology to provide supportive reminders for medication adherence has also been shown to be effective in enhancing retention and adherence.<sup>35-37</sup> Specifically, a tailored text-messaging strategy has recently shown promise with MSM.<sup>38</sup>

#### 1.2 Rationale

The purpose of this study is to develop and assess the efficacy of an integrated strategy that includes feasible and scalable interventions to identify, recruit, link to care, retain in care, and attain viral suppression among HIV-infected MSM in the US. This research is important since MSM are the most disproportionately affected population for HIV in the US, and there is an urgent need to develop innovative strategies to address this health disparity across the continuum of care. Sex between men accounted for an estimated 62% of newly identified HIV infections in the US in 2012, according to the US CDC, making enhancement of the effectiveness of engagement in care and treatment for MSM of primary importance for controlling the US domestic HIV epidemic. This study is focused on US urban MSM living with HIV infection who are not successfully virally suppressed. All MSM identified as HIV-infected and not virally suppressed will be offered linkage to care and immediate ART—an option not available in many other settings with severe epidemics among MSM. Since current HPTN sites, and concentrations of MSM in the US are primarily urban, this study will focus on urban MSM populations but may yield insights of relevance to improving outcomes for sub-urban and rural MSM in the US.

The recruitment component of this study will help refine the designs of future research and program efforts to enhance outreach, increase testing uptake and increase linkage for HIV-infected MSM who are not virally suppressed. This population includes <u>all MSM</u> with non-suppressed HIV viral loads, including men who are HIV-infected and not previously diagnosed, men who are aware of their HIV infection but not currently linked to care, and men

who may have been in care, or are currently in care, but are not successfully virally suppressed. Men in all of these groups who meet enrollment criteria will be offered enrollment in the enhanced case management intervention for linkage, retention, treatment initiation and medication adherence. DC-RDS will be assessed for its efficacy in reaching more hidden, marginalized, previously undiagnosed, and HIV-infected and not virally suppressed MSM. Future trials of enhanced treatment interventions, and of Treatment as Prevention (TasP) at community levels among MSM, will depend on the ability to reach these challenging subsets of MSM and to link them to care and treatment.

Despite clear evidence of treatment as prevention and the impact of ART on the quality and quantity of life, current data on success across the HIV treatment cascade demonstrates a need to improve both access to care and treatment adherence. Interventions to ensure MSM living with HIV and not virally suppressed are linked to and remain in care to achieve virologic control are limited and have had mixed results.<sup>39, 40</sup> Case management models, in which skilled providers facilitate HIV treatment plans to ensure appropriate and timely care are given, have been shown to be safe and improve treatment outcomes.<sup>41-43</sup> Presently, these interventions are limited to key affected populations and there is little evidence to describe the specific aspects of a case management model for linkage to care. Many studies utilizing case management models have demonstrated substantial improvements in disease outcomes, including HIV.

The Chronic Care Model (CCM) identifies essential elements of a health care system that encourage high-quality chronic disease care in a bundled approach. These elements provide the conceptual framework for the CM intervention, which is an approach to improve linkage, retention and controlled viremia in HIV-infected MSM. Tailoring of a culturally-sound case management model for MSM living with HIV and not virally suppressed may improve linkage, access, and retention in care and ultimately result in better sustained virologic control.

The use of modeling is critical to assess the potential impact of increases in the proportion of HIV-infected MSM who are successfully virally suppressed on HIV incidence in MSM networks and communities. Since this study will have an endpoint of viral suppression among HIV-infected MSM, modeling will be used to estimate the potential impact of the proposed CM intervention strategy, should it be successful, on ongoing sexual HIV transmission in selected urban US MSM networks. This ongoing MSM transmission, despite current efforts across the US, remains the largest component of incident HIV infections in the country.

Phylogenetic analysis of HIV infections among MSM could add important insights to the outreach and recruitment aims of this study. Since DC-RDS is a chain referral approach that is dependent on social and sexual networks, and participants recruit their network members for iterative recruitment waves, DC-RDS allows for the construction of network chains of referral and relatedness. As recruitment waves propagate beyond initial seeds, recruitment goes further into populations, eventually reaching significant proportions of populations with shared characteristics and who are connected through social networks. The ability to assess linkages at viral levels within these networks may provide critical insights into HIV transmission dynamics in urban MSM communities.

#### 2.0 STUDY OBJECTIVES AND DESIGN

#### 2.1 Primary Objectives

The primary objectives of the study are to:

- Assess the ability of DC-RDS to identify and recruit HIV-infected MSM in the US who are not virally suppressed.
- Compare the efficacy of the two study arms (CM intervention vs. SOC control) in achieving durable viral suppression (defined as HIV VL < 200 copies/ml) 24 months after enrollment.

# 2.2 Secondary Objectives

The secondary objectives of the study are to:

- Assess HIV prevalence and the proportion of HIV-infected men who are virally suppressed by comparing early wave (approximately 1-6) vs. later (deep) wave (approximately 7-12) DC-RDS participants.
- Compare the proportion of men in the two study arms who are virally suppressed at 3, 6 and 9, 12 and 18 months after enrollment.
- Assess linkage to care and retention in care in the two study arms by comparing the 1) proportion of men with at least one care visit within 30 days of enrollment, 2) time to the first care visit, and 3) proportion of men with at least four care visits (one in each six month interval, with at least 60 days between these visits) over the 24 months after enrollment.
- Compare the proportion of men with HIV-hepatitis C virus (HCV) co-infection in the two study arms who are linked to care (defined as one care visit within 30 days of enrollment) and who achieve (HIV) viral suppression 24 months after enrollment.
- Examine the association between baseline behavioral, socio-demographic, and clinical characteristics (including syphilis) of HIV-infected men and viral suppression status for all men screened via DC-RDS and for the men in the two study arms 24 months after enrollment.
- Compare the two study arms with respect to ART adherence at 24 months after enrollment and changes in sexual risk behavior, health care utilization, stigma, substance use and mental health from baseline to 24 months after enrollment.
- Evaluate the feasibility and scalability of the CM intervention by measuring the number of intervention contacts (e.g., text message, email, phone, in person) per participant over 24 months.
- Compare the experience of linkage to and ongoing HIV care among participants in the two study arms by conducting and analyzing exit interviews with participants and CMs.

#### 2.3 Exploratory Objectives

The exploratory objectives of the study are to:

• Use phylogenetic methods to evaluate the relationship between HIV strains in study participants. Men who were likely to have been recently infected at enrollment will be identified using a multi-assay algorithm. Evaluate the relationship of behavioral, sociodemographic, and clinical characteristics to viral networks (e.g., clusters, linked infections).

• Use laboratory assessments to characterize the study cohort and to evaluate the impacts of study interventions. These assessments may include analysis of HIV drug resistance and antiretroviral (ARV) drug use. Additional analyses may be conducted to analyze HCV strains, including phylogenetic analysis of HCV. Samples from this study may also be used to evaluate the performance of assays related to HIV and HCV infection.

# 2.4 Modeling Objective

The modeling objective of the study is to:

• Develop, calibrate, and use a mathematical model of HIV transmission among MSM in the US to assess the short and long-term population-level impact of the study strategy, and its independent CM intervention components (e.g., HIV testing, ART uptake, retention in care and viral suppression), on HIV incidence and to estimate the level of viral suppression required to reduce HIV incidence in the MSM community by 10%, 20%, 30%, and 50% over 2, 5 and 10 years, and the likelihood of and time to elimination.

# 2.5 Study Design

The overall design of this study reflects the primary goal, which is to develop and assess an integrated scalable strategy to identify, recruit, link to care, retain in care, and achieve HIV viral suppression among urban US MSM who are HIV-infected and not successfully virally suppressed. To outreach, identify and recruit HIV-infected MSM who are not virally suppressed, DC-RDS and DR will be implemented in four US cities (Atlanta, GA; Baltimore, MD; Birmingham, AL; and Boston, MA). Participating cities will have HPTN sites with evidence of high HIV burdens among MSM and interest in participating in the study. DC-RDS has been shown to be effective in reaching and identifying hard to reach subsets of MSM, including low SES, non-gay identified, and ethnic and racial minority MSM who are less likely be in HIV care and to be virally suppressed. The primary outcome of the recruitment component of the study is to assess the ability of DC-RDS to identify and recruit HIV-infected MSM in the US who are not virally suppressed.

MSM recruited through DC-RDS who meet enrollment criteria will be randomized (1:1) to one of two study arms. The intervention arm will provide a Case Manager (CM) intervention package designed to enhance linkage to care, antiretroviral treatment (ART) initiation, treatment adherence and retention in care using a case management-based intervention. The SOC control arm will provide the standard of care (SOC) for linkage to care, initiation of ART, treatment adherence and retention in care. The primary outcome of the CM intervention phase is viral suppression 24 months after enrollment.

Phylogenetic methods will be used to evaluate the relationship between viral strains in study participants and the relationship of viral networks (e.g., clusters, linked infections) to behavioral, socio-demographic, and clinical characteristics. Mathematical modeling will be performed using demographic, behavioral, and clinical data generated from this study and other sources to estimate the population-level impact of the CM intervention on HIV incidence and to estimate the level of identification, linkage, ART coverage and viral suppression that would be required to achieve a substantial reduction in HIV incidence among MSM in the US settings where the study is conducted.

#### 3.0 STUDY POPULATION

Approximately 2700 sexually active MSM (~675 in each participating city) will be recruited for HIV testing via DC-RDS and direct recruitment (DR). The study's focus is on cisgender MSM; however, transgender women who meet eligibility criteria will be included. Out of this cohort, 356 HIV-infected MSM who are not virally suppressed and meet the inclusion and exclusion criteria described below will be enrolled into the CM intervention and SOC control study arms.

#### 3.1 Inclusion Criteria

Individuals who meet all of the following criteria are eligible for study screening:

- Biological male (at birth)
- Self-report of history of anal intercourse with another man
- 16 years or older

Individuals who are eligible for screening and who meet all of the following criteria are eligible for enrollment into the CM intervention and SOC control arms:

- HIV-infected, as defined in the HPTN 078 Study-Specific Procedures (SSP) Manual
- Not virally suppressed (defined as HIV VL > 1000 copies/ml)
- Can receive HIV care at one of the participating clinics (as chosen by each site)
- No current plan to relocate in the 24 months following enrollment

#### 3.2 Exclusion Criteria

Individuals who meet any of the following criteria will be excluded from study screening:

- Unable or unwilling to provide consent/assent for study participation
- Active or previous participation in an HIV vaccine trial
- Any condition that, in the opinion of the Investigator of Record (IoR), would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Individuals who are eligible for screening, but who meet the following criteria are excluded from enrollment into the CM intervention and SOC control arms:

• Current participation in a linkage or ART adherence study

#### 3.3 Recruitment Process

DC-RDS will be used to recruit MSM into this study, to the extent possible. In this method, seeds will be identified by each site. Seeds will be the individuals who begin the recruitment chains; they will be selected to represent a range of characteristics (including ethnic and racial minority status) and because they are well-networked within the population. These seeds will undergo training to become a recruiter. They will then be given coupons with which to recruit others to the study. Seeds must meet the screening inclusion/exclusion criteria of the study and are considered study participants.

As this protocol is testing the ability of DC-RDS methodology to find HIV-positive, MSM who are not virally suppressed, DC-RDS recruitment will continue throughout the duration of the screening and enrollment period. However, DR will be used in addition to DC-RDS to fully enroll the CM intervention investigation. These new participants may be treated as seeds, if a site still needs to initiate additional recruitment chains. There will be no difference in study procedures for participants recruited via DC-RDS or DR, except that those identified via DR may or may not be treated as seeds, and thus, may or may not distribute coupons to others.

All seeds, and subsequent participant/recruiters, must not recruit anyone other than peers they know personally who are MSM. These recruits will come to the site and, if they are eligible and agree to participate, will undergo the study's screening procedures before becoming recruiters themselves. Participants will return to the clinic to be reimbursed for the coupons that were brought back to the clinic by other MSM. In addition, a post-recruitment questionnaire will be administered to characterize how many people in total were approached in the distribution of the coupons and the characteristics (e.g., age, race) of those who did and did not accept a coupon.

If necessary, more than 2700 MSM will be recruited via DC-RDS and DR to achieve the required sample size for enrollment.

#### 3.4 Co-Enrollment Guidelines

Participants will not be eligible for study participation (screening or enrollment) if they are actively or have ever been enrolled in an HIV vaccine trial, since this may affect the anti-HIV antibody profile, complicating HIV diagnosis, and use of cross-sectional methods to identify men who may have been recently infected at the time of enrollment. Participants will not be eligible for enrollment into the CM intervention and SOC control arms if they are currently participating in a linkage or ART adherence study. Once randomized, participants cannot be co-enrolled into other linkage or ART adherence studies.

# 3.5 Participant Retention

Locator information will be collected from each participant, so that they can be found if their phone number or address changes. Each site will be asked to create a retention plan to maximize the level of participation in study-required visits (follow-up visits and the final visit); however, sites will use their standard-of-care for retaining participants in clinical care throughout the study. The HPTN 078 SSP Manual will outline procedures for participants who wish to change clinics.

### 3.6 Participant Withdrawal and Early Termination

Participants may voluntarily withdraw from the study for any reason at any time. Site IoRs may, with the approval of the Protocol Chair and the Protocol statistician, withdraw participants before

their scheduled termination visit to protect their safety, and/or if participants are unable or unwilling to comply with study procedures. Participants also may be withdrawn if the study sponsors, government or regulatory authorities or site Institutional Review Boards (IRBs) terminate the study prior to its planned end date. Every reasonable effort will be made to complete a final evaluation (M24 visit procedures) of participants who terminate from the study prior to Month 24, and study staff will record the reason(s) for all withdrawals in participant study records.

# 3.7 Study Sites

Participants may be followed at participating HIV clinics in each of the four cities. All participating clinics must be able to provide the current SOC for HIV-infected MSM and be willing to provide participant information to the study team for analysis. In addition, a survey documenting standard-of-care practices will be completed for each clinic that cares for HIV-infected MSM enrolled in the study.

#### 4.0 STUDY INTERVENTION

The study CM intervention [MyLife, MyChoices, MyCare (Step 1), MyCare (Step 2), and MyHealth] is a program designed to enhance linkage, ART initiation, adherence and retention in care for MSM diagnosed with HIV. It will be administered by a trained CM and will include health care and supportive services navigation, adherence counseling, and tailored support for care engagement and treatment adherence. Table 1 and Figure 1 summarize each component, the element of the HIV care cascade it addresses and the evidence behind the CM intervention; a more complete table is included in Appendix IV.

Table 1: Tailored Case Management Intervention Components in At Risk US Populations (2005 – 2015)

| HPTN 078 Intervention<br>Component | Cascade Component | Citations |
|---|---|---|
| MyLife | <ul> <li>Linkage to care</li> <li>Engagement in care</li> <li>Retention in care</li> <li>Self-management</li> <li>Viral suppression</li> <li>Inter-personal relationship building</li> <li>Durability</li> </ul> | Hightow; 2011 <sup>48</sup><br>Quinlivan; 2013 <sup>49</sup><br>Rajabiun; 2007 <sup>50</sup><br>Yehia; 2015 <sup>51</sup> |
| MyChoices | <ul><li>Linkage to care</li><li>Engagement in care</li><li>Retention in care</li></ul> | Christopoulos; 2013 <sup>52</sup><br>Craw; 2010 <sup>53</sup> |
| MyCare (Step 1) | <ul> <li>Linkage to care</li> <li>Engagement in care</li> <li>Retention in care</li> <li>Viral suppression</li> <li>Durability</li> </ul> | Bradford; 2007 <sup>27</sup><br>Willis; 2013 <sup>47</sup> |
| MyCare (Step 2) | <ul> <li>Engagement in care</li> <li>Retention in care</li> <li>Adherence</li> <li>Viral suppression</li> <li>Inter-personal relationship building</li> <li>Durability</li> </ul> | Hayley; 2014 <sup>58</sup><br>Holtzman; 2015 <sup>59</sup><br>Naar-King; 2009 <sup>60</sup><br>Nelsen; 2013 <sup>61</sup><br>Remien; 2005 <sup>62</sup><br>Simoni; 2006 <sup>32</sup> |
| MyHealth | <ul> <li>Linkage to care</li> <li>Engagement in care</li> <li>Retention in care</li> <li>Adherence</li> <li>Self-management</li> <li>Inter-personal relationship building</li> <li>Viral suppression</li> <li>Durability</li> </ul> | Gilman; 2012 <sup>54</sup> Hightow; 2011 <sup>55</sup> Lewis; 2013 <sup>38</sup> Maulsby; 2015 <sup>56</sup> Schnall; 2015 <sup>57</sup> |




Figure 1: Relationship between the HIV Care Cascade and the CM Intervention

Based on data from: http://www.cdc.gov/hiv/pdf/research\_mmp\_stagesofcare.pdf

The CM will help each participant enrolled into the CM intervention arm to link to HIV care, initiate ART, remain adherent to medication and keeping clinical appointments. Each CM will have prior case management experience and will be trained to carry out the specified intervention aimed at improving disease management and reducing HIV viral load for patients with HIV. The CM-to-participant ratio will be approximately 1:42 over the 24-month period. As shown in Figure 2, the frequency, content and type (in person, email, phone, text message) of interactions will be driven by each patient's desire and need for support, but will minimally follow the schedule of events (see Appendix I). All CM-participant interactions will be documented (frequency and duration) to assess the feasibility and scalability of the CM intervention. To ensure uniformity and fidelity of the intervention across sites, each CM will undergo a standardized, comprehensive training program, and each mandatory session (at required study visits) will be audio recorded and a small percentage will be assessed against a standard counselling index, as described in the HPTN 078 SSP Manual.

Figure 2: Overview of CM-Administered Study Intervention



Note: Some participants may choose to meet in person with the CM on a very frequent basis (e.g. weekly); these visits will be documented, however, such visits are not mandatory and there are no required study procedures during them.

This CM-led model builds upon the existing CDC-endorsed Comprehensive Risk Counseling and Services for Persons with HIV<sup>63</sup>, which focuses on the prevention of HIV transmission. The model combines aspect of clinical care coordination to include; a) recruitment and engagement (MyLife); b) inventory of available resources (MyChoices); c) patient navigation to clinical care (MyCare (Step 1)); d) adherence counseling (MyCare (Step 2); e) retention and follow-up (MyHealth).

The approach of the CM follows an approach similar to HPTN 073 in the use of a self-determination theoretical approach, which hypothesizes that reestablishing autonomy is a key element for long-term engagement in care for some patients. <sup>49</sup> Additionally, the Gelberg-Andersen Behavioral Model for vulnerable populations <sup>64</sup> will be used to identify enabling, predisposing and need variables that impact adherence and retention in care, which has been effectively demonstrated in women living with HIV, but not in an MSM group. <sup>65</sup> The role of the CM within each of the five components is described below.

Participants enrolled into the SOC control arm will be provided with the existing programs for referral to HIV treatment and support services without additional CM coordination.

# 4.1 Linkage to Care and ART Initiation (MyLife, MyChoices, MyCare (Step 1))

#### 4.1.1 Engagement (MyLife)

The MyLife component is the first step of the CM intervention as developing a therapeutic or interpersonal relationship with the participant is the paramount first step. Engaging with the participant is an effective strategy that has been shown to improve retention. Fart of this engagement process is to attempt to understand the participant's state of mind after the HIV diagnosis and address any HIV-related questions they may have. It may become necessary to end the first session here depending on the individuals needs related to their diagnosis. This session will include an HIV counseling intervention about the new diagnosis and an overview of the case management model in support of the patient. The CM will be taught motivational interviewing skills to facilitate participant engagement into clinical practice.

After the initial question-answer period, the CM will seek to understand the predisposing, enabling and health needs of the participant.<sup>64</sup> A standardized instrument will be utilized to elicit this information from the patient. Once these data are available, the CM will discuss and assist the participant to develop an individually-tailored plan that is designed utilizing self-determination theory. Self-determination theory is anchored by three core components: (1) autonomy support-provision of evidence-based health guidance and supporting the participant-endorsement of the plan they believe best meets their needs and fits within their life circumstance; (2) competence support-expression of belief in the participants' ability to implement their self-endorsed plan and provision of guidance for acquiring the necessary skills and resources for successful implementation; and (3) relational support-expression/demonstration of genuine care and concern for the participant's successful implementation of the plan (e.g., follow-up phone/text check-ins). These three components are theorized to facilitate the adoption and maintenance of health behaviors. A comprehensive training program on the use of this model will be provided to all CMs.

#### 4.1.2 Inventory of Available Resources (MyChoices)

MyChoices will involve a discussion of resources available to meet the participants stated healthcare needs. The CM will have a comprehensive listing of available HIV, substance abuse, mental health, and other available resources to discuss with the participant. The CM will provide guidance on options that work within the delineated plan and make modifications based on the participant's needs and review of the available resources.

#### 4.1.3 Patient Navigation to Clinical Care (MyCare (Step 1))

MyCare (Step 1) supports the decision to initiate HIV care and will include motivational interviewing activities to coach the client toward seeking and initiating care. Once care decisions have been made by the participant, the CM will offer to facilitate entry into the care facility selected by the patient. This will include the establishment of necessary appointments, facilitation of paperwork and registration materials, pre-clinical laboratory evaluations, evaluation of provider options within the clinical site as well as introductions of the clinical team through either website review, phone calls, or a clinic visit with onsite team prior to the first visit. All participants will be encouraged to initiate (or re-initiate) ART in consultation with their healthcare provider.


# 4.2 Adherence Counseling (MyCare (Step 2))

In conjunction with ART initiation, the CM will deliver evidence-based adherence counseling, which will be modeled after Life Steps<sup>31</sup>, a single-session intervention that is grounded in cognitive-behavioral principles that are at the core of several successful ART adherence interventions. <sup>25, 32, 62, 66</sup> The adherence counseling will address basic education about HIV and ART, planning and problem-solving for accessing and maintaining a steady supply of medication, formulation of a daily medication schedule, cues for pill-taking, coping with side effects and/or other patient concerns, developing a plan to mitigate side effects, and responses to slips in adherence. This counseling will be provided face-to-face prior to, at the time of, or in the very early stage of ART initiation. Participants will be encouraged to bring a support partner to the adherence counseling sessions, if they so desire, which has been shown to be effective for long-term medication adherence. <sup>62, 66, 67</sup> The counseling intervention allows for tailoring to the participants specific needs, as well as additional counseling sessions, if needed. MyCare (Step 2) adds to this evidence-based approach by recognizing that adherence to treatment is a personal choice that is grounded in a variety of behavioral and psychosocial domains. Intention to adhere to treatment will be added as part of the MyCare (Step 2) component. <sup>61</sup>

# 4.3 Communication, Retention and Follow-up (MyHealth)

MyHealth is based on the premise that all patients engaged in self-management and supportive strategies will feel more empowered to take ownership of their own healthcare needs. In addition, there is accumulated evidence for the acceptability and preference for two-way text messaging for adherence support among diverse populations, including MSM. 35-38 As such, tailored communication support will be offered to facilitate ongoing adherence. The CM will work with each participant to determine their desire for supportive adherence reminders, their preferred method of communication (text message, email or phone call), and the frequency and schedule for these messages. In this way, the participant is being empowered to take the lead with recommendations and guidance from the CM. This type of messaging is interactive in that it allows for a response from participants, in case a participant needs additional information or assistance. The frequency and content of these communications may change over the course of the intervention, depending on the needs of the participant.

#### 5.0 STUDY PROCEDURES

An overview of the study visits and procedures is presented in Appendix I. Additional information is provided below on visit-specific study procedures. Detailed instructions to guide and standardize all study procedures across sites will be provided in the SSP Manual.

#### 5.1 Screening Visits

There are several algorithms for screening visits (see HPTN 078 SSP Manual). The timing of screening activities will vary between algorithms, but all screening activities described below will be completed for each algorithm. Additionally, re-screening for eligibility is allowed under certain circumstances (see HPTN 078 SSP Manual).

All individuals will be consented for screening procedures, which include the provision of contact information, completion of several questionnaires (see Appendix II) and samples collected for laboratory assessments. All participants will undergo HIV screening (via one Food and Drug Administration (FDA)-approved HIV rapid test [either oral fluid or finger stick or whole blood], self-report, or clinic record) and have blood drawn for HCV and syphilis testing. For those who report being previously diagnosed with HIV infection, have HIV infection documented in a clinic record, or have a reactive rapid HIV test, additional blood will be collected for HIV confirmatory testing (see HPTN 078 SSP Manual), HIV viral load and CD4+ cell count. In addition, pre- and post-test HIV counseling and HIV/sexually transmitted infection (STI) risk reduction counseling will be provided to all participants, as appropriate. Participants will also be assessed for social impacts that may have occurred during the recruitment process.

Participants who participate in DC-RDS will also be given instructions about the recruitment process and coupons for distribution. Additionally, if applicable at later visits, a post-recruitment questionnaire will be administered to DC-RDS participants who have distributed their coupons.

All participants, regardless of eligibility, may be provided with their test results by phone or in-person, per site standards. If the HCV and/or syphilis test are positive, participants will be referred for care via site standards. Participants who are eligible and willing to enroll may be provided with their test results in-person on the day of their enrollment visit.

# 5.1.1 Procedures for Participants Who are Determined to be HIV-Uninfected

Participants who are determined to be HIV-uninfected (see HPTN 078 SSP Manual) will be given information on HIV prevention, including current information about pre-exposure prophylaxis (PrEP) and post-exposure prophylaxis (PEP). These participants are not eligible for enrollment into the CM intervention or SOC control arms.

#### 5.1.2 Procedures for Participants Who are Confirmed to be HIV-Infected

Participants who are confirmed to be HIV-infected (see HPTN 078 SSP Manual) will be screened for participation in the intervention, and, if eligible, will be invited to be enrolled into the CM intervention or SOC control arms. If an individual is eligible for randomization, but chooses not to participate further in the study, they will be referred to local HIV care facilities.

# 5.1.3 Procedures for Participants Whose HIV Status is Inconclusive

Participants whose HIV status is not clear after their last screening visit will be referred to a local care provider for further evaluation and follow-up. If such a participant is later confirmed to be HIV-infected, they may be re-assessed for eligibility (see HPTN 078 SSP Manual).

#### 5.2 Enrollment Visit (M0)

The Enrollment Visit will take place as soon as participants are determined to be eligible. During this visit, participants will be consented for enrollment and randomized to either the CM intervention or SOC control arm. Participants will be asked to sign a release of medical information, their locator information will be confirmed, they will be asked to complete a questionnaire (see Appendix II), and they will have blood drawn for plasma storage. All participants will be offered HIV testing for their partners. Depending on the results of the partners' HIV test results, partners will be referred to appropriate HIV care services or other HIV-related studies. [Note: partner testing will be done outside of the study and results will not be recorded.] In addition, the intervention will begin at this visit for those randomized to the CM intervention arm, and, if appropriate, ART may be initiated at this visit. (Note that ART is not provided by the study, nor prescribed by the CM.)

#### **5.3** Tailored Communication

Once an individual is enrolled into the CM intervention arm, they will decide how much, if any, text message, email or phone reminders they would like to receive to support ART adherence. These reminders will be tailored to the needs of the participant so that they are effective, while maintaining privacy. The CM will facilitate the distribution of these messages and respond to requests for assistance via these two-way modes of communication. This tailored communication to support ART adherence will not be offered to participants in the SOC control arm.

# **5.4** Monthly Contact

The CM will contact each participant randomized to the CM intervention arm on a monthly basis to confirm their locator information, to check-in with the participant regarding HIV and ART management, and to collect any social impacts due to study participation. Participants may choose this contact to be in person or by text message, email or phone call. No monthly contact will be made with participants in the SOC control arm.

#### 5.5 Follow-up Visits (M3, M6, M9, M12, M18)

Follow-up Visits will take place at Months 3, 6, 9, 12 and 18 for all participants (CM intervention and SOC control arms). During these face-to-face visits, locator information will be confirmed, social impacts will be collected, partner HIV testing will be offered, HIV viral load and CD4 cell count testing will be conducted, and plasma will be stored. For those randomized to the CM intervention arm, the intervention will be implemented by the CM.

# 5.6 Final Visit (M24)

The Final Visit will take place at Month 24. This visit will be identical to a Follow-up Visit, except that blood will be collected for syphilis testing and questionnaires will be administered (see Appendix II). An exit interview will also be conducted or scheduled with all participants. If the syphilis test is positive, participants will be given their test results and referred for care via site standards. An exit interview will be conducted with each CM after they complete the final visit for their last participant.

#### 5.7 Data Collection on ART Initiation and Visit Attendance

Information about ART initiation, if it takes place during study follow-up, and overall visit attendance will be collected from all participants' medical records.

#### 5.8 **Questionnaires**

#### **5.8.1** Participant Questionnaires

Questionnaires in the following domains will be administered over the course of the study: demographic; PrEP/PEP/ART use history; HIV testing history; sexual matrix module/sexual risk behavior; health care utilization; engagement in the lesbian, gay, bisexual and transgender (LGBT) community; post recruitment questions; medication adherence; stigma; substance abuse; and mental health. The schedule for these questionnaires is provided in Appendix II. When possible, the domain questionnaires will be adapted from recent MSM-focused HPTN studies such as HPTN 061 and 073 to allow cross comparison. Additionally, validated questions/scales from the literature will be used to gain information in domains that are vital to understanding the impact of the study design and intervention. Information on the focus of each domain is provided below:

- **Demographic:** Data collected in this domain will include information such as age, gender, marital status, education, annual income, race/ethnicity and health insurance status.
- **PEP/PrEP/ART:** Information collected in this domain will focus on actual behaviors and use of PEP/PrEP/ART in the last 12 months. Daily and intermittent use of PrEP in the community will also be evaluated.
- **HIV testing history:** The HIV testing history domain will document how many times the participant has been tested for HIV in the past year and the month and year of the most recent HIV test. In addition, this domain will document whether the participant received the results and if so, the result of the test.
- **Sexual matrix module/Sexual risk behavior:** Information collected within these domains will include information on number of partners, frequency and types of sexual acts, and geography of the sexual experiences. This information will help identify sexual exposures inside and outside the defined community. The questions in this domain will be adapted from both HPTN 061 and HPTN 073 as well as the Berry sexual activity matrix.<sup>68, 69</sup>
- **Health care utilization:** Information collected in this domain will include information on health care utilization and services and assess engagement at baseline. Trust between the clinician and patient will also be evaluated. Information in this domain will also be collected

at the final visit to assess any supplemental services that have been accessed outside the study.

- Engagement in the LGBT community: Information collected in this domain will include information on how well people are engaged and connected in the LGBT community. This domain will supplement the post recruitment questions and allow the team to evaluate the effectiveness of DC-RDS in finding those connected and individuals that are hidden in the community. This may reveal any association with the likelihood of being undiagnosed.
- **Post recruitment questions:** Information collected in this domain will focus on evaluating the effectiveness of DC-RDS and recruitment strategies by participants.<sup>70, 71</sup>
- **Stigma:** Information collected in this domain will be very focused on self-stigma (internalized homo-negativity) and HIV stigma (with consideration of impact on HIV testing and adherence). This questionnaire domain is being adapted from Herek et al 1997.<sup>72</sup>
- Substance abuse and mental health: Information collected in this section will focus on depression, post-traumatic stress disorder, anxiety and substance abuse. These assessments will be brief screeners that the case manager can use to intervene or provide referrals. The Substance Abuse/Mental Illness Symptoms Screener (SAMISS)<sup>73, 74</sup> will be the primary source for this domain.
- **Medication adherence:** This domain will be self-reported medication adherence. A three-item scale developed by Wilson et al, <sup>75</sup> which has recently been shown to be correlated with HIV viral load outcomes across different populations, will be used.
- Exit Interview: A questionnaire and a semi-structured qualitative interview will be administered to participants asking them to describe their experiences with linkage-to-care, adherence and the CM intervention; information will be collected from both arms about outside interventions/care. Such exit interviews will also be conducted with the CMs, with the questions tailored for their role in the study.

# 5.8.2 Site Questionnaires

Site questionnaires will be administered to each site providing care to HPTN 078 enrolled participants to document their standard of care. These surveys will be administered annually to capture sites' normal procedures throughout the duration of the study.

#### 6.0 SAFETY MONITORING AND ADVERSE EVENT REPORTING

# 6.1 Safety Monitoring

As this study only involves low-risk activities (recruitment activities; testing for HIV, HCV, and syphilis; questionnaires; support for linkage-to-care, care engagement and ART adherence) and contains no biomedical intervention or clinical care (ART prescription or other medical treatment), standard adverse event reporting will not be undertaken. The study team will collect and report all social impacts that are brought to the attention of study staff members. Research staff will be trained to recognize and report social impacts as well as provided with referrals for counseling and social service support, if necessary. Reports of social impacts will be reviewed quarterly or more often, if indicated, and reported to the DAIDS Medical Officer together with any actions that are taken. Social impacts will be summarized and reported to appropriate Institutional Review Boards (IRB)(s) on an annual basis.

Confidential HIV and STI surveillance reporting will be done according to local regulations. Participants will be reminded of these requirements via the Informed Consent Form.

# 6.2 Social Impact Reporting

It is possible that participants' involvement in the study could become known to others, and that a social impact may result (i.e., because participants could be perceived as being HIV-infected or at "high risk" for HIV infection). For example, participants could be treated unfairly, or could have problems being accepted by their families and/or communities. A social impact that is reported by the participant and judged by the Investigator of Record (IoR) or designee to be serious or unexpected will be reported to the responsible site's IRBs at least annually, or according to their individual requirements. Social impacts will be collected and reported on case report forms (CRFs) during regular visits. In the event that a participant reports a social impact, every effort will be made by study staff to provide appropriate care and counseling to the participant as necessary, and/or referral to appropriate resources for the safety of the participant. While maintaining participant confidentiality, study sites may engage their Community Advisory Board (CAB) in exploring the social context surrounding instances of social impacts, to minimize the potential occurrence of such a harm.

#### 7.0 STATISTICAL CONSIDERATIONS

#### 7.1 Review of Study Design

This study is designed to i) evaluate the utility of DC-RDS for finding HIV-infected MSM who are not virally suppressed, and ii) assess the efficacy of an CM intervention package for linking HIV-infected MSM to care and, ultimately, achieving viral suppression. Approximately 2700 MSM will be identified and recruited (see Sections 7.2.1 and 7.6.1 for definition of recruitment) using DC-RDS and DR strategies in four cities (~675 per city). We expect that approximately 378 of these will be HIV-infected MSM who are not virally suppressed and that 356 of these will be willing to participate. These 356 individuals will be randomized to the CM intervention and SOC control study arms of the study. The CM intervention arm will provide a package designed to enhance linkage to care, ART initiation, treatment adherence, and retention in care. The intervention will be delivered by a trained CM. The SOC control arm will provide the SOC for linkage to care, initiation of ART, and treatment. The primary outcome of the study is viral suppression 24 months after enrollment.

# 7.2 Endpoints

#### 7.2.1 Primary Endpoints

Consistent with the primary study objective to assess the ability of DC-RDS to identify and recruit HIV-infected MSM in the US who are not virally suppressed, the following endpoints will be assessed:

- HIV status at screening for each MSM recruited by DC-RDS
- HIV viral load at screening for each HIV-infected MSM recruited by DC-RDS

Consistent with the primary study objective to compare the efficacy of the two study arms (CM intervention vs. SOC) in achieving viral suppression (defined as HIV VL <200 copies/ml) 24 months after enrollment, the following endpoint will be assessed:

• HIV viral load at 24 months after enrollment

# 7.2.2 Secondary Endpoints

Consistent with the secondary study objective to assess HIV prevalence and the proportion of men who are virally suppressed by comparing early wave (approximately 1-6) vs. later (deep) wave (approximately 7-12) DC-RDS participants, the following endpoint will be assessed:

• Date and wave of recruitment for each man recruited by DC-RDS

Consistent with the secondary study objective to compare the proportion of men in the two study arms who are virally suppressed (defined as HIV VL <200 copies/ml) at 3, 6, 9, 12 and 18 months after randomization the following endpoints will be assessed:

• HIV viral load at 3, 6, 9, 12 and 18 months after enrollment

Consistent with the secondary study objective to compare the proportion of men in the two study arms who are linked to care and retained in care the following endpoints will be assessed:

Number and time of all care visits from randomization through the end of 24 month follow-up

Consistent with the secondary study objective to compare the proportion of men with HIV-HCV co-infection who are linked to care and who achieve HIV viral suppression 24 months after enrollment between the two study arms the following endpoint will be assessed:

- HCV status at baseline
- HIV viral load at 24 months after enrollment

Consistent with the secondary study objective to examine the association between baseline behavioral, socio-demographic, and clinical characteristics of HIV-infected men and viral suppression status for all men screened via DC-RDS and for the men in the two study arms 24 months after enrollment the following endpoints will be assessed:

- Self-reported sexual risk behavior (number of male sexual partners, episodes of unprotected anal intercourse [UAI], characteristics of 3 most recent partners) at baseline using a standardized assessment tool
- Age, education, and other socio-demographic measures at baseline
- CD4, HIV viral load and syphilis status at baseline

Consistent with the secondary study objective to compare ART adherence at 24 months and changes in sexual risk behavior, health care utilization, stigma, substance use and mental health between the two study arms over 24 months, the following endpoint(s) will be assessed:

- Self-reported sexual risk behavior (number of male sexual partners, episodes of UAI, characteristics of 3 most recent partners) at baseline and 24 months using a standardized assessment tool
- ART adherence at 24 months
- Health care utilization at baseline and 24 months using a standardized assessment tool
- Stigma at baseline and 24 months using a standardized assessment tool
- Substance use at baseline and 24 months using a standardized assessment tool
- Mental health at baseline and 24 months using a standardized assessment tool

Consistent with the secondary study objective to evaluate the feasibility and scalability of the CM intervention package, the following endpoint(s) will be assessed:

• Number of contacts (text message, email, phone, in person) for each participant randomized to the CM intervention arm over follow-up

Consistent with the secondary study objective to compare the experience of linkage to and ongoing HIV care among participants in the two study arms, the following endpoint(s) will be assessed:

- Satisfaction with the CM intervention components, as measured on a Likert scale during a standardized exit interview
- Usefulness of the CM intervention components, as measured on a Likert scale during a standardized exit interview
- Open-ended questions for process evaluation

# 7.2.3 Exploratory Endpoints

- Consistent with the exploratory study objective to use phylogenetic methods to evaluate the relationship between behavioral, socio-demographic, and clinical characteristics and viral networks (e.g., clusters, linked infections).
  - The phylogenetic relationship between HIV sequences

Consistent with the exploratory study objective to use laboratory assessments to characterize the study cohort and to evaluate the impacts of study interventions, the following endpoint(s) may be assessed:

 Laboratory measures that may include HIV drug resistance, detection of ARV drugs and other assessments

# 7.3 Accrual, Follow-up and Sample Size

We will recruit approximately 2700 men via DC-RDS and DR. We expect that 20% (540) will be HIV-infected MSM and that 70% of those (378) will not be suppressed. These 378 individuals form the pool of individuals eligible for enrollment and randomization. If necessary, more than 2700 MSM will be recruited via both methods to achieve the required sample size for enrollment.

We expect that 40% of the MSM randomized to the SOC control arm will be linked to care and 70% of those linked to care will be suppressed by 24 months following enrollment. We expect that almost none of those not linked to care will be suppressed. Thus, overall, we expect about 28% of the MSM in the SOC control condition will be suppressed at 24 months. In the CM intervention arm we expect to raise the linkage rate to at least 55% and the suppression rate, among those linked, to 85%. Thus, we expect that at least 46% of the MSM in the CM intervention arm will be suppressed at 24 months. Table 2 shows the required sample size for an individually randomized trial with 90% power, assuming 10% lost-to-follow-up per year, for various effect sizes. For our target effect size of risk difference of 18% points, we require 356 MSM.

Table 2. Number needed to be randomized to the CM intervention or SOC control to have 90% power to detect the indicated difference in proportion of those virally suppressed at 24 months, assuming  $\alpha = 0.05$  (two-tailed), power = 90%, loss to follow-up = 10%/year (overall retention of 80% at the end of 2 years).

| Difference in proportion suppressed at 24 months between arms <sup>1</sup> | 0.12 | 0.18 | 0.24 |
|---|---|---|---|
| Number randomized | 780 | 356 | 190 |

<sup>&</sup>lt;sup>1</sup>Valid for SOC control group viral suppression rates between  $\sim 30 - 50\%$ .

Table 3 shows the precision of estimates of i) awareness of HIV-infected status and ii) viral suppression among those who are HIV-infected, based on the DC-RDS sample.

Table 3. Precision for estimating the indicated proportions, assuming 20% of DC-RDS recruits are HIV-infected

| Number recruited via DC-RDS | Expected number HIV-infected | Awareness of HIV-infected status (expected proportion = 0.20) | Virally suppressed at enrollment among HIV-infected (expected = 0.25) |
|---|---|---|---|
| 2000 | 400 | +/-0.039 | +/-0.042 |
| 1500 | 300 | +/-0.045 | +/-0.049 |
| 1000 | 200 | +/-0.055 | +/-0.060 |

# 7.4 Random Assignment

HIV-infected MSM who are recruited by the DC-RDS or DR, are eligible and agree to participate in the study will be randomized in a 1:1 ratio to the CM intervention and SOC control arms using randomly-permuted blocks, stratified by site.

The randomization scheme will be generated and maintained by the HPTN SDMC. Additional details regarding the process of randomization will be included in the SSP Manual.

#### 7.5 Blinding

Participants and study investigators will not be blinded to the randomization assignments.

#### 7.6 Data Analysis

#### 7.6.1 Primary Analysis

To assess the ability of DC-RDS to recruit HIV-infected MSM who are not virally suppressed we will measure the proportion of the men that are recruited by DC-RDS (where recruitment is defined as providing a blood draw for HIV and HIV viral load testing) who are HIV-infected and not virally suppressed. An estimate and a 95% confidence interval (CI) based on RDS methods<sup>76</sup> will be reported. MSM recruited via other methods will not be included in this analysis.

Among the HIV-infected MSM who are enrolled and randomized we will compare the rates of viral suppression (defined as HIV VL <200 copies/ml) at 24 months after enrollment. The absolute difference in the probability of viral suppression between the CM intervention and SOC control arms and a 95% CI will be reported. A chi-squared test with a two-sided alpha level of 0.05 will be used for testing the hypothesis:

Ho: No difference in suppression between arms

Ha: Difference in suppression between arms

The analysis will follow the intent to treat principle. If a participant drops out prior to 24 months, their viral suppression status at last study assessment will be used in the analysis. A sensitivity analysis will be conducted to evaluate the effect of different assumptions about the viral suppression status of those who drop out.
As a secondary analysis, we will repeat the above for the subgroup of randomized participants who are HCV seropositive at baseline.

# 7.6.2 Secondary Analysis

We will divide the MSM who are recruited into early and later waves of DC-RDS (the definition of "early" and "late" will be included in the statistical analysis plan). We will use a two sample test of proportions (with standard errors adjusted for RDS sampling;<sup>76</sup>) to compare i) the proportion HIV-infected and ii) the proportion HIV-infected and not suppressed, between the early and later recruits. MSM recruited via other methods will not be included in this analysis. A two-sided alpha level of 0.05 will be used for hypothesis testing.

We will also repeat the analysis of HIV viral suppression (described in Section 7.6.1) at 3, 6, 9, 12 and 18 months of follow-up. As in the primary analysis, viral suppression status at last study assessment will be used for participants who drop out prior to a time point. Chi-squared tests with a two-sided alpha level of 0.05 will be used at each time point.

Among the HIV-infected MSM who are enrolled and randomized, we will compare the rates of linkage to care (defined as at least one care visit within 30 days of enrollment) between the CM intervention and SOC control arm. Any randomized participant who drops out of the study prior to 30 days will be counted as "not linked" for the purpose of this analysis. The absolute difference in the probability of linkage between the CM intervention and SOC control arms and a 95% CI will be reported. A chi-squared test with a two-sided alpha level of 0.05 will be used for hypothesis testing. Similarly, we will use a Cox regression model to compare time to first linkage visit between the two study arms. A hazard ratio and 95% CI will be reported. Both analyses will follow the intent to treat principle.

We will also compare the proportion of MSM who are retained in care (defined as at least four care visits [one in each six-month interval, with at least 60 days between these visits] over the 24 months after enrollment) between the CM intervention and SOC control arm. Any randomized participant who drops out of the study without at least two care visits as defined above will be counted as "not retained" for the purpose of this analysis. The absolute difference in the probability of retention between the CM intervention and SOC control arms and a 95% CI will be reported. A chi-squared test with a two-sided alpha level of 0.05 will be used for hypothesis testing. The analysis will follow the intent to treat principle.

We will build a multiple logistic regression model to examine the associations between viral suppression at 24 months (outcome) and various demographic characteristics, sexual risk behaviors and clinical characteristics. Further details will be provided in a separate Statistical Analysis Plan.

Additional analyses will examine the effect of the CM intervention on various sexual risk behavior, ART adherence, stigma, health care use, substance use and mental health measures over the 24 month follow-up. The general approach to these analyses will be to build a regression model (linear, log, or logistic, whichever is appropriate for the scale of the measure) that uses the 24 month value of the measure as the outcome (or most recent assessment for participants that drop out prior to 24 months) and includes the baseline value of the measure (except for ART adherence, where no baseline value is available) and CM intervention arm as covariates. The coefficient of the CM intervention arm covariate will be used to quantify the CM intervention effect. An estimate of the CM intervention effect and a 95% CI will be provided for each outcome. Further details will be provided in a separate Statistical Analysis Plan.

Among those randomized to the CM intervention arm we will measure the number of contacts (text message, email, phone, in person) per participant over follow-up. Summary statistics (mean, median, interquartile range, etc.), standardized by the number of months in follow-up, will be provided.

We will summarize the distribution of responses on satisfaction with and usefulness of the CM intervention components from the exit interviews using means, medians and interquartile ranges.

# 7.6.3 Qualitative Analysis

We will conduct qualitative analysis of all open-ended process evaluation data by coding and analyzing the qualitative data utilizing a qualitative software package for systematic data management (e.g., NVivo) to evaluate participants' and CMs' reactions, preferences and recommendations for treatment interventions.

# 7.6.4 Exploratory Analysis

Phylogenetic trees will be built using HIV sequences from study participants and other relevant sequences (e.g., controls). If viral networks are identified (e.g., clusters, linked infections), we will evaluate the relationship of behavioral, socio-demographic, and clinical characteristics to viral networks.

If other exploratory laboratory assessments are performed (e.g., drug resistance, ARV drug use, HCV phylogenetics), the HPTN Laboratory Center (LC) will identify specific endpoints for analysis.

## 8.0 HUMAN SUBJECTS CONSIDERATIONS

#### 8.1 Ethical Review

This protocol and the template informed consent form(s) contained in Appendix III will be reviewed and approved by the HPTN Scientific Review Committee (SRC) and NIAID Prevention Science Review Committee (PSRC) with respect to scientific content and compliance with applicable research and human subjects regulations.

The protocol, site-specific informed consent form, participant education and recruitment materials, and other requested documents — and any subsequent modifications —will also be reviewed and approved by the ethical review bodies responsible for oversight of research conducted at each study site.

Subsequent to initial review and approval, the responsible IRBs will review the protocol at least annually. The Investigators of Record will make safety and progress reports to the IRBs at least annually, and within three months of study termination or completion. These reports will include the total number of participants enrolled in the study, the number of participants who completed the study, all changes in the research activity, and all unanticipated problems involving risks to human subjects or others. Study sites are responsible for the submission of continuing review documentation to the DAIDS Protocol Registration Office, in accordance with the current DAIDS Protocol Registration Policy and Procedure Manual.

#### 8.2 Informed Consent

Written informed consent will be obtained from each study participant prior to conducting study-related procedures. Each study site is responsible for developing a study informed consent form for local use, based on the templates in Appendix III, which describe the purpose of the study, the procedures to be followed, and the risks and benefits of participation, in accordance with all applicable regulations. Based on local IRB approval and state law, sites may seek a waiver of parental consent for either the DC-RDS activities alone or both the DC-RDS and CM activities. However, only sites that are granted a waiver of parental consent for the DC-RDS activities will be allowed to screen minors (16 and 17 year olds).

Participants will document their provision of informed consent by signing the informed consent forms. (Further details regarding DAIDS requirements for documenting the informed consent process are provided in the DAIDS Standard Operating Procedure for Source Documentation.)

All participants will be offered a copy of their informed consent forms.

## 8.3 Incentives

Pending IRB approval, participants may be compensated for their time and effort for study-required activities, or reimbursed for travel to study-required visits or time away from work for study-required activities. Site-specific reimbursement amounts will be specified in the study informed consent forms.

## 8.4 Confidentiality

All study-related information will be stored securely at each study site. All participant information will be stored in locked file cabinets in areas with access limited to study staff. All

laboratory specimens, reports, study data collection, process, and administrative forms will be identified by a coded number only to maintain participant confidentiality. All records that contain names or other personal identifiers, such as locator forms and informed consent forms, will be stored separately from study records identified by code number. All local databases will be secured with password-protected access systems. Forms, lists, logbooks, appointment books, and any other listings that link participant identification (ID) numbers to other identifying information will be stored in a separate, locked file in an area with limited access.

Participant's study information will not be released without the written permission of the participant, except as necessary for monitoring by NIAID and its contractors; representatives of the HPTN Leadership and Operations Center (LOC), SDMC, or HPTN LC; Office for Human Research Protections (OHRP) or other government and regulatory authorities; or site IRBs.

The HPTN will obtain a Certificate of Confidentiality from the U.S. Department of Health and Human Services that will be applicable for this study. Sites may register under the Certificate through the HPTN LOC once they have obtained local IRB approval for the study. This Certificate protects study staff from being compelled to disclose study-related information by any Federal, State or local civil, criminal, administrative, legislative, or other body.

## 8.5 Communicable Disease Reporting Requirements

Study staff will comply with all applicable local requirements to report communicable diseases identified among study participants to local health authorities. Participants will be made aware of all reporting requirements during the study informed consent process.

## 8.6 Study Discontinuation

The study also may be discontinued at any time by NIAID, the HPTN, OHRP or other government or regulatory authorities, or site IRBs.

## 9.0 LABORATORY SPECIMENS AND BIOHARDS CONTAINMENT

Laboratory procedures are described below and in Appendix I.

# 9.1 Local Laboratory Specimens

Specimens will be collected for testing at the local laboratory. Laboratory evaluations/procedures will include:

- HIV testing (see SSP Manual)
- Syphilis testing
- HCV testing (see SSP Manual)
- CD4 cell count testing
- HIV viral load testing
- Plasma storage

Local laboratories and clinics where testing is performed must be certified under the Continuous Laboratory Improvement Amendment (CLIA-certified) or must be in possession of a CLIA Waiver. Additional local and State guidelines must also be followed.

Each study site will adhere to standards of good clinical laboratory practice, and local standard operating procedures for specimen management including proper collection, processing, labeling, transport, and storage of specimens to the local laboratories. Specimen storage at the local laboratory will be documented using the HPTN Laboratory Data Management System (LDMS) as described in the SSP Manual.

# 9.2 LC Specimens

Specimens will be collected for testing at the HPTN LC. Laboratory evaluations and procedures will include:

- HIV quality assurance (QA) testing
- Other testing\*

\*Stored plasma will be used for QA testing and other assessments at the HPTN LC. This may include cross-sectional incidence testing (to identify participants who are recently infected at Enrollment). Stored samples will also be used for phylogenetic analysis. Other assessments that may be performed include ARV drug testing; HIV resistance testing; characterization of HIV and HCV and the host response to viral infection. Samples collected in the study may also be used to evaluate assays related to HIV and HCV infection. In some cases, testing will be performed at a commercial laboratory or another laboratory designated by the HPTN LC. These assessments will be performed retrospectively; results will not be returned to study sites or participants (with the possible exception of HIV diagnostic testing, if results obtained at the HPTN LC differ from site results).

# 9.3 Quality Control and Quality Assurance Procedures

HPTN LC staff will conduct periodic visits to each site to assess the implementation of on-site laboratory quality control (QC) procedures, including proper maintenance of laboratory testing equipment and use of appropriate reagents. HPTN LC staff will follow up directly with site staff to resolve any QC or QA problems identified through proficiency testing and/or on-site assessments.

# 9.4 QC for HIV Diagnostic Testing

The HPTN LC will perform HIV diagnostic testing for QC. Algorithms for HIV diagnostic testing are provided in the SSP Manual.

# 9.5 Phylogenetic Analysis

Phylogenetic methods will be used to explore the relationship between viruses from study participants. HIV sequencing will be performed at the HPTN LC or another laboratory designated by the HPTN LC. HIV sequencing will be performed by bulk (population) sequencing; next generation/deep sequencing may also be performed. The HPTN LC will determine the methods used for phylogenetic analysis (e.g., the HIV genomic regions analyzed, use of local and other control sequences, methodology used for data analysis).

# 9.6 Specimen Storage and Possible Future Research Testing

Study site staff will store all plasma specimens collected in this study at for at least three years after the end of the study (completion of the last study visit). In addition, study participants will be asked to provide written informed consent for their plasma specimens to be stored after the end of the study for possible future testing related to HIV and HCV infection, evaluation of laboratory assays relevant to the study objectives, and other assessments. The specimens of participants who do not consent to long-term storage and additional testing will be destroyed after all protocol-related testing has been completed; sample destruction must be coordinated with the HPTN LC and HPTN SDMC.

# 9.7 Biohazard Containment

As the transmission of HIV and other blood-borne pathogens can occur through contact with contaminated needles, blood, and blood products, appropriate blood and secretion precautions will be employed by all personnel in the drawing of blood and shipping and handling of all specimens for this study, as currently recommended by the US CDC. All infectious specimens will be transported in accordance with US regulations (42 Code of Federal Regulations [CFR] 72).

## 9.8 Resistance Testing at Local Laboratories.

HIV resistance testing may be performed at local laboratories for clinical management using locally-available resistance test methods. Study specimens may not be used for this testing; additional specimens must be collected for this testing. Resistance testing may also be performed at the HPTN LC or a laboratory designated by the HPTN LC using stored specimens; results of this testing will not be returned to study sites or study participants.

## 10.0 MODELING COMPONENT

#### 10.1 Background and Prior Research

Mathematical models of HIV transmission are widely used to understand the dynamics of HIV transmission, to assess the population-level impact of HIV prevention and treatment interventions and to inform policy decisions. 77 They are also increasingly and innovatively being used at different stages of the clinical trial process: to inform product development, to inform the design of optimal combination prevention, to inform the design and conduct of large community-based clinical trials, and to interpret and help generalize results to the wider population.<sup>78</sup> Models of HIV transmission amongst MSM have been used to estimate the impact of role segregation (taking only the insertive or receptive role in anal intercourse), 79-81 and serosorting (having anal sex only with MSM of the same HIV status), 82,83 which both lead to lower overall HIV prevalence. Models have also been used to understand the racial disparities in HIV prevalence seen amongst MSM in the US, 84 which are related to preferential mixing by race, and differences in access to care and treatment. Models have been used to estimate the impact of pre-exposure prophylaxis for MSM in the US85 and Peru,86 informed by effectiveness estimates from the iPrEx trial of PrEP for MSM. Modelling has also been used to estimate the likely impact of increasing HIV testing and treatment amongst MSM. For example, modeling has been used to predict a moderate impact of increased testing frequency alone for MSM, 15, 87 to estimate the impact of behavior change following HIV testing<sup>88</sup> and to predict a more substantial impact from increased testing coupled with immediate ART treatment for MSM. 15, 89, 90

In the current study, models will be used to estimate the likely population level impact on HIV transmission of the increased rates of identification of HIV-infected non-virally suppressed MSM and the increased level of viral suppression achieved in the trial, and to estimate the effect of the different trial components, which aim to increase the identification of unsuppressed HIV-infected MSM and increase linkage to care, ART initiation and retention in care.

#### 10.2 Rationale

Mathematical modelling will be used to translate the results of the study and estimate the potential population-level impact of the tested CM intervention on HIV, since the trial does not include HIV incidence as an endpoint and will measure the impact of the CM intervention at an individual rather than a community level. Rather than measuring the impact of the CM intervention upon HIV incidence, the first main objective of the study is to measure the success of the DC-RDS strategy in finding MSM who are not virally suppressed (primary objective), while also capturing useful information about the risk profile (behavioral, socio-demographic and clinical) of the population reached and retained at different stages of the treatment cascade (secondary objective). The second primary objective of the study is to measure the impact of the CM intervention upon the proportion of MSM achieving viral suppression after 24 months (primary objective), and the time to viral suppression (secondary objective), as well as collecting data on intermediate steps including the proportion linked to care and remaining engaged in care (secondary objective).

Given the focus on treatment outcomes and the endpoint of viral suppression, and the fact that the CM intervention can influence multiple outcomes on the causal HIV prevention pathway among HIV-infected MSM (e.g. increased initiation and retention in treatment, changes in sexual behavior), it is difficult to understand the prevention potential of the individual-level CM intervention on population-level HIV incidence based on the trial results alone. Mathematical models are needed to translate the results of the CM intervention components implemented in this


study into estimates of the potential population-level impact of the combined CM intervention package on future HIV acquisition and transmission, taking into account the specific risk profile of those adopting the CM intervention and the existing epidemiological and prevention contexts where the interventions are taking place.

Models can also be used to estimate the level of treatment-as-prevention efforts required to reduce HIV incidence at the population level by a substantial amount as rapidly as possible, and to assess whether the results of this trial in terms of CM intervention uptake, retention, adherence, and the risk profile of the population reached and responding favorably to the CM intervention warrant roll-out of the CM intervention to the wider MSM population.

## 10.3 Model Population and Setting

The modelled population will be all sexually active MSM (both HIV-infected and HIV-uninfected) in each of the four different sites included in the trial.

#### 10.4 Main Model Outcomes

The main model outcomes include the following:

- Predicted population-level reduction in incidence and prevalence achieved by the CM intervention, and by individual components of the CM intervention (HIV testing, ART uptake, retention in care and viral suppression) over 2, 5 and 10 years at each site.
- Predicted preventable fraction (PF): The fraction of new HIV infections averted by a given CM intervention package, or its independent components, over a fixed time period
- Estimated level of viral suppression required to reduce HIV incidence at each site by 10%, 20%, 30%, and 50% over 2, 5 and 10 years.
- Estimates of whether or not the CM intervention would be likely to result in HIV elimination (HIV incidence less than one new HIV infection per 1000 people per year<sup>91</sup>) at each site, and the time taken to reach this elimination threshold, both with achieved levels of viral suppression, and for the different levels of viral suppression required to meet incidence reduction targets.
- Population attributable fraction (PAF): The contribution of different risk groups or risk factors to HIV transmission over different time periods.

# 10.5 Modeling Stages

We will develop and analyze a dynamical, deterministic compartmental model of sexual HIV transmission and HIV prevention among MSM in different US settings, and use it to estimate the impact of the CM intervention at the population level.

For each setting, the modeling study will include a number of stages:

- Model development and coding
- Model parameterization
- Model calibration and fitting to HIV prevalence and incidence data from various site specific sources
- Model analysis: estimation of CM intervention impact, including uncertainty and sensitivity analysis

More details about the different stages are given in the following sections.

## 10.5.1 Model Development and Coding

The proposed model is a dynamic, deterministic compartmental model which describes HIV transmission via anal sex between and among different risk groups of MSM, as well as rates of HIV progression and levels of testing and treatment over time. Within the model, the MSM population will be divided into different categories stratified by age, race, sexual risk activity (e.g. rate of partner acquisition, frequency of sex acts)<sup>92, 93</sup> and sexual role behavior (exclusively insertive, exclusively receptive, or versatile in anal sex) (Figure 3).<sup>80, 94</sup>

Figure 3: Behavioral Groups and Sexual Mixing in the Model.



MSM are divided into different groups relating to sexual role behavior (exclusively insertive, exclusively receptive, or versatile in anal sex), age, race and sexual risk activity. MSM in each of these groups may be uninfected with HIV (gray), infected and not virally suppressed (red; highly infectious), or infected, treated and virally suppressed (green; reduced infectiousness). Sexual mixing between these groups will be informed by data on mixing patterns by age, race, sexual risk and sexual role. As ART coverage increases (i.e. the proportion of sexual partners on ART increases), HIV viral load will decrease (viral suppression increases) and so HIV incidence will decrease.

In the model, HIV infection and progression will be modelled as a number of discrete stages through which MSM move – susceptible (uninfected), acute HIV infection (stage 1), chronic HIV infection, divided into three stages (stages 2-4), and AIDS (stage 5; Figure 4). This staging allows the model to reflect changes in infectivity, CD4 levels and symptoms which occur as a function of time since infection, and to capture historical changes in the timing of treatment initiation. HIV-infected MSM with acute infection or AIDS will have increased infectivity, and those on ART and virally suppressed will have reduced infectivity (Figures 3 and 4). HIV-infected MSM may move between different categories reflecting their testing and treatment status, including those unaware of their HIV positive status, those tested, linked into pre-ART care, those on ART and partially or fully virally suppressed and those who are lost to follow-up, have discontinued ART and those living with HIV who have never been tested. This last category contains individuals who may also initiate ART when they present with symptoms (Figure 4).



Figure 4: Infection and Treatment States.

MSM in the model are divided into separate categories by infection and treatment status. Infected MSM are divided by infection stage, with the chronic phase subdivided into several stages (reflecting CD4 levels when untreated) to allow more accurate timing of AIDS, appearance of symptoms and ART initiation and modelling historical increases in treatment which was based on CD4 levels. MSM on ART have greatly reduced infectivity when they are virally suppressed. The level of infectiousness is indicated in pink/red/green. MSM start ART either due to presenting symptoms or following testing.

The force of HIV infection (or per capita HIV incidence rate) for susceptible MSM will be estimated (following calibration, details below) based upon the frequency and type of sex acts (insertive/receptive) they have, as well as condom use with different types of partner (main, casual and commercial), their circumcision status, PrEP and PEP use, who their sexual partners are likely to be (based upon mixing preferences related to age, race, sexual risk activity and serostatus and data on the proportion of sexual partners resident inside and outside of the study community), and levels of HIV prevalence and ART use among those partners (Figure 5). To capture the impact of other STIs upon HIV transmission risk, syphilis prevalence measured at baseline will be used together with published estimates of the increased risk of HIV transmission in the presence of syphilis to estimate associated increases in HIV transmission in each setting, assuming stable syphilis prevalence. The final model structure will depend upon the site-specific data available (from the trial and other complementary sources) to determine parameters and also upon important identified sources of heterogeneity.

Figure 5: Force of Infection.



This figure summarizes the different factors which contribute to the force of infection (per capita incidence rate), including characteristics of the susceptible MSM and of their sexual partners.

The model will incorporate the effects over time of past and existing interventions (e.g., increases in condom and ART use), and future interventions (the CM intervention and standard of care, including associated levels of linkage to care, ART initiation and adherence and retention in care), upon HIV susceptibility, transmissibility and rate of disease progression. Changes in levels of HIV testing will also be represented, as will documented changes in sexual behavior (including number and type of partners and sexual mixing patterns).

The model will consist of coupled nonlinear ordinary differential equations and will be coded with a flexible programming language (e.g. C++).

#### 10.5.2 Model Parameterization

The data required to inform model parameters and calibrate the model cover five main domains: demography, sexual behavior, natural history of HIV, intervention, and epidemiological HIV data. This information should ideally be obtained from representative samples of the population. We will use data from the trial (which may need to be standardized to reflect the wider MSM population, and to account for the recruitment process), and we will also comprehensively review and make use of other relevant sources of data such as HIV surveillance data, the published literature, systematic reviews and official reports. The trial will provide data to inform the modelling of future interventions, including data on the demography, sexual behavior, prior HIV testing, HIV prevalence, viral status, and ART use of those recruited through DC-RDS. The trial will also provide estimates of the proportion of people linking to and retained in care, initiating ART and achieving viral suppression, with and without the CM intervention package. In addition, the trial will provide data on the demographic and risk profiles of those retained at each stage of the HIV care cascade. Complementary data from other sources will be needed to inform modelling of past behavior and interventions and to characterize the wider MSM population at each site (including demographic, sexual behavior and HIV testing data). Other data will also be required to model the progression of HIV and effectiveness of different interventions, and to capture historical changes in behavior and ART coverage. Likely sources of data to inform the CM intervention and standard of care scenarios are summarized in Table 4; the final data sources used may vary depending upon the exact sites used for the trial.

Table 4. Model parameters and likely data sources

| Data<br>Domain | Parameters | Trial Data Used | Other Data Used |
|---|---|---|---|
| Demography | Age composition, natural death rates, MSM population size, migration | RDS-derived estimates of population size, age, mobility data, data on whether sex partners are resident inside/outside the community | Age composition: overall for national sample (NHBS); Natural death rates: National Vital Statistics reports; total population size: US Census data; Proportion of people reporting same-sex sexual activity: National Survey of Family Growth (NSFG) |
| Sexual<br>Behavior | Number and type of male anal sex partners (per unit time), frequency of insertive and receptive anal sex with different partners, preference for partners by age, race, HIV status and sexual activity, role behavior, condom use with different partners. Changes in these behaviors over time | Number of partners and sex acts, role behavior, condom use at baseline (RDS + CM intervention cohort) and after 24 months (CM intervention cohort only), partner characteristics at baseline (RDS + CM intervention cohort) | Number of main and casual partners last year: Overall estimate from CDC NHBS surveys for MSM 2005, 2008, 2011, 2014; overall number of male partners last year: NSFG, national estimate; condom use at last sex act: overall estimate from NHBS surveys 2005, 2008, 2011, 2014; levels of consistent condom use: NHBS individual sites 2005, 2008, 2011, 2014; role behavior <sup>92</sup> |
| Natural<br>History of<br>HIV | Duration, probability of infection per sex act (by role), infectivity by HIV viral load | (no trial data will be used) | Duration of different stages of infection: European cohort studies <sup>96</sup> Relative infectiousness of different stages of infection: published analyses <sup>97</sup> Probability of infection per anal sex act: published literature and existing systematic reviews <sup>97-99</sup> Infectivity by HIV viral load: <sup>15, 100-102</sup> |

| Data<br>Domain | Parameters | Trial Data Used | Other Data Used |
|---|---|---|---|
| CM<br>intervention<br>and SOC | Rates of HIV testing, linkage to care, ART initiation, viral suppression; PrEP and PEP use; changes in these over time and differences between study arms. Retention in care and ART adherence. Loss to follow- up. Effectiveness of male circumcision, condoms, ART, PrEP in reducing infectiousness | Current levels PrEP and PEP use, HIV testing, ART coverage in RDS sample; levels of HIV testing post-recruitment among RDS sample; linkage to care, ART initiation, adherence, retention in care, viral suppression for each arm of the trial, by risk group, and loss to follow-up. | Testing: CDC NHBS surveys for MSM (for NHBS sites) Linkage to care, ART initiation, viral suppression: CDC MMWR reports Published literature and systematic reviews on effectiveness of male circumcision, 103 condoms, 104, 105 ART, PrEP |
| HIV<br>Epidemiology | HIV prevalence and incidence, changes over time, distribution of transmission by sources of infection; distribution among treated and untreated | HIV prevalence in RDS population HIV incidence estimates using laboratory assays (if conducted) Phylogenetic analysis Baseline distribution of treated and untreated HIV-infected; both suppressed and unsurpassed | Prevalence: CDC NHBS<br>surveys for MSM 2005,<br>2008, 2011, 2014 (for<br>NHBS sites)<br>Incidence: CDC estimates<br>for MSM 2005 (selected<br>NHBS sites), cohort data<br>where available |

MMWR, Morbidity and Mortality Weekly Report; NHBS, National HIV Behavioral Surveillance; NSFG, National Survey of Family Growth.

For each model parameter, a most likely value and a range of plausible values (a priori range) will be obtained.

# 10.5.3 Model Calibration and Fitting

The model, including past and current levels of interventions, will be calibrated to available HIV prevalence and incidence data over time (which is representative of the sites modelled) within a Bayesian framework where *a priori* information on the key parameters from available data sources is updated through a comparison of the model simulations and epidemiological HIV data. The parameter ranges constructed in the model parameterization stage will be exhaustively sampled and explored at the calibration stage, using state of the art fitting methods previously used 107-109 in order to identify multiple parameter sets that agree with the epidemiological HIV data (HIV prevalence and incidence), producing a set of model predictions which reflect HIV patterns by risk group in the target population while taking into account uncertainty in parameter assumptions. This set of simulations will form our baseline scenario and baseline parameter sets. As per standard procedure in modelling studies, 94, 95, 107, 108, 110 this calibrated set of simulations will also produce the necessary baseline estimates of population level HIV incidence required to subsequently be able to assess the impact of scaling up future interventions.

## 10.5.4 Model Analysis

The calibrated model for each site will be used to conduct the following analyses: (1) assess the population level impact of the overall study strategy on HIV incidence and prevalence, and the preventable fraction of HIV infections averted; (2) assess the population level impact of the individual components of the CM intervention (including HIV testing, ART uptake, retention in care, viral suppression) on HIV incidence and prevalence and the preventable fraction of HIV infections averted by these individual components; (3) estimate the level of viral suppression required to reduce HIV incidence at each site by 10%, 20%, 30%, and 50% over 2, 5 and 10 years; (4) estimate the likelihood of and time taken to reach HIV elimination; (5) estimate the PAF for different risk groups, the stage in the cascade of care and the risk factors over different time periods; (6) uncertainty and sensitivity analyses.

## 10.5.4.1Overall CM Intervention Impact

The model will be run for each site under two alternative scenarios, standard of care (baseline) and CM intervention, with levels of testing, linkage, ART initiation and retention, and viral suppression going into the future informed by the levels measured in each arm of the trial (table 1). Predicted overall CM intervention impact will be determined by comparing the predicted cumulative HIV incidence, HIV incidence rate and HIV prevalence in the CM intervention and baseline scenarios over 2, 5 and 10 years, with all trial components included in the intervention arm. This will yield estimates of the impact of the total CM intervention package on population-level HIV incidence and prevalence, and the preventable fraction PF(dt) of HIV infections. In these analyses we will take into account differences in CM intervention coverage and uptake by risk group. Each modelling outcome will be presented as the mean, median and uncertainty range (95% percentiles of the model predictions based on the multiple posterior parameter sets).

# 10.5.4.2 Impact of Individual CM Intervention Components

We will then use the models to estimate the impact of the observed independent CM intervention components, by running additional model scenarios in which only some of the CM intervention components (increased rates of HIV testing, increased linkage, ART uptake, retention in treatment and viral suppression) are included, and comparing these with the baseline model in the same way as for the full CM intervention model, above, to estimate the reduction in incidence and prevalence and the PF associated with each CM intervention component and combination of components. Each modelling outcome will be presented as the mean, median and uncertainty range (95% percentiles of the model predictions based on the multiple posterior parameter sets).

## 10.5.4.3 Required Viral Suppression to Achieve Incidence Reduction Targets

We will also use the models to estimate the level of viral suppression and associated CM intervention efforts that need to be achieved in order to reduce HIV incidence in the MSM community by 10%, 20%, 30%, and 50% over 2, 5 and 10 years.

#### 10.5.4.4 HIV Elimination

We will estimate whether HIV is predicted to be eliminated if the CM intervention were carried on into the future for each site, both with achieved levels of viral suppression, and for the different levels of viral suppression required to meet the incidence reduction targets (10%, 20%, 30%, and 50% reduction over 2, 5 and 10 years). Elimination is defined as HIV incidence going below one new HIV infection per 1000 people per year. 91 Where elimination is predicted, we will estimate the predicted time taken to reach the elimination threshold.

Each study outcome will be presented as the mean, median and uncertainty range (95% percentiles of the model predictions based on the multiple posterior parameter sets).

## 10.5.4.5 Population Attributable Fraction (PAF)

We will determine the main drivers of HIV acquisition and transmission in the MSM populations studied by calculating the short and long term transmission PAF. <sup>111, 112</sup> The PAF(dt) will be derived by comparing the number of new infections using two defined risk parameters: 1) assuming that the given risk factor increases risk of HIV acquisition or transmission or the relevant risk behavior; 2) assuming no increase in risk associated with the factor under study. The key risk groups for whom we will calculate PAFs will be: sexual role groups (insertive or receptive, versatile), untested MSM, and HIV-infected MSM who not virally suppressed.

# 10.5.4.6 Uncertainty and Sensitivity Analyses

We will conduct an uncertainty analysis using the multiple calibrated simulations to assess the influence of key epidemiological and intervention factors/parameters (in CM intervention and SOC control arms) on impact predictions (using a technique such as partial rank correlation), and determine under which conditions a CM intervention will have the largest impact (using techniques such as regression trees analysis).

We will conduct a sensitivity analysis to determine the influence on the impact estimates (incidence and prevalence reduction and PF) of key parameters such as the evolution of the SOC over time, and determine a threshold of high sensitivity where impact is considerably reduced.

## 11.0 ADMINISTRATIVE PROCEDURES

## 11.1 Protocol Registration

Initial Registration of the protocol by the DAIDS Protocol Registration Office (PRO) is required prior to implementation of this protocol. As part of this process, each site must have the protocol and protocol informed consent form(s) approved, as appropriate, by their local IRB/ethics committee (EC) and any other applicable regulatory entity. Upon receiving final approval, sites will submit all required protocol registration documents to the DAIDS PRO at the Regulatory Support Center (RSC). The DAIDS PRO will review the submitted protocol registration packet to ensure that all of the required documents have been received. In the case of Initial Registration, site-specific informed consent forms (ICFs) will be reviewed and approved by the DAIDS PRO. Sites will receive an Initial Registration Notification from the DAIDS PRO that indicates successful completion of the protocol registration process. A copy of the Initial Registration Notification should be retained in the site's regulatory files.

Following Initial Registration, any full protocol amendments require submission of a protocol registration packet to the DAIDS PRO as described above; however, the DAIDS PRO will not review and approve site-specific ICFs. Sites will receive a Registration Notification when the DAIDS PRO receives a complete registration packet.

For additional information on the protocol registration process and specific documents required for initial and amendment registrations, refer to the current version of the DAIDS Protocol Registration Manual, which can be found at http://rsc.tech-res.com/protocolregistration/.

## 11.2 Study Activation

Pending successful protocol registration and submission of all required documents, the HPTN LOC staff will "activate" a site. Study implementation may not be initiated until a study activation notice is provided to the site by the HPTN LOC. In addition, if study "activation" is determined to be necessary for any subsequent amendments, study implementation may not be initiated until a study activation notice is provided to the site by the HPTN LOC.

## 11.3 Study Coordination

Study implementation will be directed by this protocol as well as the SSP Manual. The SSP Manual will outline procedures for conducting study visits; data and forms processing; social harm assessment, management and reporting; and other study operations.

Study CRFs and other study instruments will be developed by the protocol team and HPTN SDMC. Data will be transferred to the HPTN SDMC for data entry, cleaning, reporting and analysis. Quality control reports and queries will be generated and distributed to the study sites on a routine schedule for verification and resolution.

Close coordination between protocol team members will be necessary to track study progress, respond to queries about proper study implementation, and address other issues in a timely manner. Rates of accrual, adherence, follow-up, and social harm incidence will be monitored closely by the team as well as the HPTN Study Monitoring Committee (SMC). The Protocol Chair, DAIDS Medical Officer, Protocol Biostatistician, SDMC Project Manager, and HPTN LOC representatives will address issues related to study eligibility and social harm management

and reporting as needed to assure consistent case management, documentation, and information-sharing across sites.

# 11.4 Study Monitoring

On-site study monitoring will be performed in accordance with DAIDS policies. Study monitors will visit the site to:

- Verify compliance with human subjects and other research regulations and guidelines;
- Assess adherence to the study protocol, study-specific procedures manual, and local counseling practices; and
- Confirm the quality and accuracy of information collected at the study site and entered into the study database.

Site investigators will allow study monitors to inspect study facilities and documentation (e.g., informed consent forms, clinic and laboratory records, other source documents, CRFs), as well as observe the performance of study procedures. Investigators also will allow inspection of all study-related documentation by authorized representatives of the HPTN LOC, HPTN SDMC, HPTN LC, NIAID, site IRBs/ECs, and US regulatory authorities (OHRP). A site visit log will be maintained at each study site to document all visits.

## 11.5 Protocol Compliance

The study will be conducted in full compliance with the protocol. The protocol will not be amended without prior written approval by the Protocol Chair and DAIDS Medical Officer. All protocol amendments must be submitted to and approved by the relevant IRB(s) and the DAIDS RSC prior to implementing the amendment.

#### 11.6 Investigator's Records

All site Investigators of Record (IoR) will be responsible for maintaining, and storing in a secure manner, complete, accurate, and current study records throughout the study. Under the US Department of Health and Human Services (HHS) regulations, the IoR is required to retain all study records relating to research for at least three [3] years after completion of the research, or longer if needed to comply with local regulations. Completion of a clinical research study occurs when the following activities have been completed:

- All research-related interventions or interactions with human subjects;
- All protocol-required data collection of identifiable private information described in the IRB/EC-approved research plan;
- All analysis of identifiable private information described in the IRB/EC-approved research plan;
- Primary analysis of either identifiable private or de-identified information.

Study records include administrative documentation — including protocol registration documents and all reports and correspondence relating to the study — as well as documentation related to

each participant screened and/or enrolled in the study — including informed consent forms, locator forms, CRFs, notations of all contacts with the participant, and all other source documents.

# 11.7 Use of Information and Publications

Publication of the results of this study will be governed by the HPTN Manual of Operations. Any presentation, abstract, or manuscript will be submitted to the HPTN Manuscript Review Committee and DAIDS for review prior to submission.

## 12.0 REFERENCES

- 1. Beyrer C, Sullivan P, Sanchez J, et al. The increase in global HIV epidemics in MSM. *AIDS* 2013; **27**(17): 2665-78.
- 2. Centers for Disease Control and Prevention. HIV Surveillance Report, Volume 23. 2011. <a href="http://www.cdc.gov/hiv/pdf/statistics\_2011\_hiv\_surveillance\_report\_vol\_23.pdf">http://www.cdc.gov/hiv/pdf/statistics\_2011\_hiv\_surveillance\_report\_vol\_23.pdf</a> (accessed August 29 2014).
- 3. Millett GA, Peterson JL, Flores SA, et al. Comparisons of disparities and risks of HIV infection in black and other men who have sex with men in Canada, UK, and USA: a meta-analysis. *Lancet* 2012; **380**(9839): 341-8.
- 4. Centers for Disease Control and Prevention. HIV Among Gay and Bisexual Men. 2015. <a href="http://www.cdc.gov/nchhstp/newsroom/docs/CDC-MSM-508.pdf">http://www.cdc.gov/nchhstp/newsroom/docs/CDC-MSM-508.pdf</a> (accessed September 12 2015).
- 5. Koblin BA, Mayer KH, Eshleman SH, et al. Correlates of HIV acquisition in a cohort of Black men who have sex with men in the United States: HIV prevention trials network (HPTN) 061. *PloS one* 2013; **8**(7): e70413.
- 6. Bradley H, Hall HI, Wolitski RJ, et al. Vital Signs: HIV diagnosis, care, and treatment among persons living with HIV--United States, 2011. *MMWR Morbidity and mortality weekly report* 2014; **63**(47): 1113-7.
- 7. Paz-Bailey G, Miller W, Shiraishi RW, Jacobson JO, Abimbola TO, Chen SY. Reaching men who have sex with men: a comparison of respondent-driven sampling and timelocation sampling in Guatemala City. *AIDS and behavior* 2013; **17**(9): 3081-90.
- 8. Wei C, McFarland W, Colfax GN, Fuqua V, Raymond HF. Reaching black men who have sex with men: a comparison between respondent-driven sampling and time-location sampling. *Sexually transmitted infections* 2012; **88**(8): 622-6.
- 9. Fuqua V, Chen YH, Packer T, et al. Using social networks to reach Black MSM for HIV testing and linkage to care. *AIDS and behavior* 2012; **16**(2): 256-65.
- 10. Millett GA, Ding H, Marks G, et al. Mistaken assumptions and missed opportunities: correlates of undiagnosed HIV infection among black and Latino men who have sex with men. *J Acquir Immune Defic Syndr* 2011; **58**(1): 64-71.
- 11. Baral SD, Ketende S, Schwartz S, et al. Evaluating Respondent-Driven Sampling as an Implementation Tool for Universal Coverage of Antiretroviral Studies Among Men Who Have Sex With Men Living With HIV. *J Acquir Immune Defic Syndr* in press.
- 12. Coombs A, McFarland W, Ick T, Fuqua V, Buchbinder SP, Fuchs JD. Long-chain peer referral to recruit black MSM and black transgender women for an HIV vaccine efficacy trial. *J Acquir Immune Defic Syndr* 2014; **66**(4): e94-7.
- 13. Das M, Chu PL, Santos GM, et al. Decreases in community viral load are accompanied by reductions in new HIV infections in San Francisco. *PloS one* 2010; **5**(6): e11068.
- 14. Frange P, Meyer L, Deveau C, et al. Recent HIV-1 infection contributes to the viral diffusion over the French territory with a recent increasing frequency. *PloS one* 2012; **7**(2): e31695.
- 15. Phillips AN, Cambiano V, Nakagawa F, et al. Increased HIV incidence in men who have sex with men despite high levels of ART-induced viral suppression: analysis of an extensively documented epidemic. *PloS one* 2013; **8**(2): e55312.

- 16. Cohen MS, Chen YQ, McCauley M, et al. Prevention of HIV-1 infection with early antiretroviral therapy. *The New England journal of medicine* 2011; **365**(6): 493-505.
- 17. Rosenberg ES, Rothenberg RB, Kleinbaum DG, Stephenson RB, Sullivan PS. The implications of respondent concurrency on sex partner risk in a national, web-based study of men who have sex with men in the United States. *J Acquir Immune Defic Syndr* 2013; **63**(4): 514-21.
- 18. Christopoulos KA, Das M, Colfax GN. Linkage and retention in HIV care among men who have sex with men in the United States. *Clinical infectious diseases : an official publication of the Infectious Diseases Society of America* 2011; **52 Suppl 2**: S214-22.
- 19. Hightow-Weidman LB, Jones K, Phillips G, 2nd, Wohl A, Giordano TP. Baseline clinical characteristics, antiretroviral therapy use, and viral load suppression among HIV-positive young men of color who have sex with men. *AIDS patient care and STDs* 2011; **25 Suppl** 1: S9-14.
- 20. Magnus M, Jones K, Phillips G, 2nd, et al. Characteristics associated with retention among African American and Latino adolescent HIV-positive men: results from the outreach, care, and prevention to engage HIV-seropositive young MSM of color special project of national significance initiative. *J Acquir Immune Defic Syndr* 2010; **53**(4): 529-36.
- 21. Wohl AR, Galvan FH, Myers HF, et al. Do social support, stress, disclosure and stigma influence retention in HIV care for Latino and African American men who have sex with men and women? *AIDS and behavior* 2011; **15**(6): 1098-110.
- 22. Robbins RN, Spector AY, Mellins CA, Remien RH. Optimizing ART Adherence: Update for HIV Treatment and Prevention. *Current HIV/AIDS reports* 2014; **11**(4): 423-33.
- 23. Nachega JB, Uthman OA, Mills EJ, Quinn TC. Adherence to Antiretroviral Therapy for the Success of Emerging Interventions to Prevent HIV Transmission: A Wake up Call. *Journal of AIDS & clinical research* 2013; **2012**(Suppl 4).
- 24. Simoni JM, Amico KR, Smith L, Nelson K. Antiretroviral adherence interventions: translating research findings to the real world clinic. *Current HIV/AIDS reports* 2010; **7**(1): 44-51.
- 25. Thompson MA, Mugavero MJ, Amico KR, et al. Guidelines for improving entry into and retention in care and antiretroviral adherence for persons with HIV: evidence-based recommendations from an International Association of Physicians in AIDS Care panel. *Annals of internal medicine* 2012; **156**(11): 817-33, W-284, W-5, W-6, W-7, W-8, W-9, W-90, W-91, W-92, W-93, W-94.
- 26. Craig C, Eby D, Whittington J, Institute for Healthcare Improvement. Care Coordination Model: Better care at lower cost for people with multiple health and social needs. 2011. <a href="https://www.IHI.org">www.IHI.org</a> (accessed July 10 2014).
- 27. Bradford JB, Coleman S, Cunningham W. HIV System Navigation: an emerging model to improve HIV care access. *AIDS patient care and STDs* 2007; **21 Suppl 1**: S49-58.
- 28. Craw JA, Gardner LI, Marks G, et al. Brief strengths-based case management promotes entry into HIV medical care: results of the antiretroviral treatment access study-II. *J Acquir Immune Defic Syndr* 2008; **47**(5): 597-606.
- 29. Johnson D, Polansky M, Matosky M, Teti M. Psychosocial factors associated with successful transition into HIV case management for those without primary care in an urban area. *AIDS and behavior* 2010; **14**(2): 459-68.

- 30. Chaiyachati KH, Ogbuoji O, Price M, Suthar AB, Negussie EK, Barnighausen T. Interventions to improve adherence to antiretroviral therapy: a rapid systematic review. *AIDS* 2014; **28 Suppl 2**: S187-204.
- 31. Safren SA, Otto MW, Worth JL. Life-steps: Applying cognitive behavioral therapy to HIV medication adherence. *Cognitive and Behavioral Practice* 1999; **6**: 332–41.
- 32. Simoni JM, Pearson CR, Pantalone DW, Marks G, Crepaz N. Efficacy of interventions in improving highly active antiretroviral therapy adherence and HIV-1 RNA viral load. A meta-analytic review of randomized controlled trials. *J Acquir Immune Defic Syndr* 2006; **43 Suppl 1**: S23-35.
- 33. DiMatteo MR. Social support and patient adherence to medical treatment: a meta-analysis. Health psychology: official journal of the Division of Health Psychology, American Psychological Association 2004; 23(2): 207-18.
- 34. Safren SA, O'Cleirigh CM, Skeer M, Elsesser SA, Mayer KH. Project enhance: a randomized controlled trial of an individualized HIV prevention intervention for HIV-infected men who have sex with men conducted in a primary care setting. *Health psychology: official journal of the Division of Health Psychology, American Psychological Association* 2013; **32**(2): 171-9.
- 35. Huang D, Sangthong R, McNeil E, Chongsuvivatwong V, Zheng W, Yang X. Effects of a Phone Call Intervention to Promote Adherence to Antiretroviral Therapy and Quality of Life of HIV/AIDS Patients in Baoshan, China: A Randomized Controlled Trial. *AIDS research and treatment* 2013; **2013**: 580974.
- 36. Lester RT, Ritvo P, Mills EJ, et al. Effects of a mobile phone short message service on antiretroviral treatment adherence in Kenya (WelTel Kenya1): a randomised trial. *Lancet* 2010; **376**(9755): 1838-45.
- 37. Sidney K, Antony J, Rodrigues R, et al. Supporting patient adherence to antiretrovirals using mobile phone reminders: patient responses from South India. *AIDS care* 2012; **24**(5): 612-7.
- 38. Lewis MA, Uhrig JD, Bann CM, et al. Tailored text messaging intervention for HIV adherence: a proof-of-concept study. *Health psychology: official journal of the Division of Health Psychology, American Psychological Association* 2013; **32**(3): 248-53.
- 39. Vital signs: HIV prevention through care and treatment--United States. *MMWR Morbidity and mortality weekly report* 2011; **60**(47): 1618-23.
- 40. Gardner EM, McLees MP, Steiner JF, Del Rio C, Burman WJ. The spectrum of engagement in HIV care and its relevance to test-and-treat strategies for prevention of HIV infection. *Clinical infectious diseases : an official publication of the Infectious Diseases Society of America* 2011; **52**(6): 793-800.
- 41. Anaya HD, Hoang T, Golden JF, et al. Improving HIV screening and receipt of results by nurse-initiated streamlined counseling and rapid testing. *Journal of general internal medicine* 2008; **23**(6): 800-7.
- 42. Andersen MD, Smereck GA, Hockman EM, Ross DJ, Ground KJ. Nurses decrease barriers to health care by "hyperlinking" multiple-diagnosed women living with HIV/AIDS into care. *The Journal of the Association of Nurses in AIDS Care : JANAC* 1999; **10**(2): 55-65.
- 43. Schumann A, Nyamathi A, Stein JA. HIV risk reduction in a nurse case-managed TB and HIV intervention among homeless adults. *Journal of health psychology* 2007; **12**(5): 833-43.

- 44. Brennan A, Browne JP, Horgan M. A systematic review of health service interventions to improve linkage with or retention in HIV care. *AIDS care* 2014; **26**(7): 804-12.
- 45. Gallant JE, Adimora AA, Carmichael JK, et al. Essential components of effective HIV care: a policy paper of the HIV Medicine Association of the Infectious Diseases Society of America and the Ryan White Medical Providers Coalition. *Clinical infectious diseases: an official publication of the Infectious Diseases Society of America* 2011; **53**(11): 1043-50.
- 46. Pasricha A, Deinstadt RT, Moher D, Killoran A, Rourke SB, Kendall CE. Chronic Care Model Decision Support and Clinical Information Systems interventions for people living with HIV: a systematic review. *Journal of general internal medicine* 2013; **28**(1): 127-35.
- 47. Willis S, Castel AD, Ahmed T, Olejemeh C, Frison L, Kharfen M. Linkage, engagement, and viral suppression rates among HIV-infected persons receiving care at medical case management programs in Washington, DC. *J Acquir Immune Defic Syndr* 2013; **64 Suppl** 1: S33-41.
- 48. Hightow-Weidman LB, Smith JC, Valera E, Matthews DD, Lyons P. Keeping them in "STYLE": finding, linking, and retaining young HIV-positive black and Latino men who have sex with men in care. *AIDS patient care and STDs* 2011; **25**(1): 37-45.
- 49. Quinlivan EB, Messer LC, Adimora AA, et al. Experiences with HIV testing, entry, and engagement in care by HIV-infected women of color, and the need for autonomy, competency, and relatedness. *AIDS patient care and STDs* 2013; **27**(7): 408-15.
- 50. Rajabiun S, Mallinson RK, McCoy K, et al. "Getting me back on track": the role of outreach interventions in engaging and retaining people living with HIV/AIDS in medical care. *AIDS patient care and STDs* 2007; **21 Suppl** 1: S20-9.
- 51. Yehia BR, Ketner E, Momplaisir F, et al. Location of HIV diagnosis impacts linkage to medical care. *J Acquir Immune Defic Syndr* 2015; **68**(3): 304-9.
- 52. Christopoulos KA, Massey AD, Lopez AM, et al. "Taking a half day at a time:" patient perspectives and the HIV engagement in care continuum. *AIDS patient care and STDs* 2013; **27**(4): 223-30.
- 53. Craw J, Gardner L, Rossman A, et al. Structural factors and best practices in implementing a linkage to HIV care program using the ARTAS model. *BMC health services research* 2010; **10**: 246.
- 54. Gilman B, Hidalgo J, Thomas C, Au M, Hargreaves M. Linkages to care for newly diagnosed individuals who test HIV positive in nonprimary care settings. *AIDS patient care and STDs* 2012; **26**(3): 132-40.
- 55. Hightow-Weidman LB, Jones K, Wohl AR, et al. Early linkage and retention in care: findings from the outreach, linkage, and retention in care initiative among young men of color who have sex with men. *AIDS patient care and STDs* 2011; **25 Suppl 1**: S31-8.
- 56. Maulsby C, The Positive Charge Intervention T, Charles V, et al. Positive Charge: Filling the Gaps in the U.S. HIV Continuum of Care. *AIDS and behavior* 2015.
- 57. Schnall R, Bakken S, Rojas M, Travers J, Carballo-Dieguez A. mHealth Technology as a Persuasive Tool for Treatment, Care and Management of Persons Living with HIV. *AIDS and behavior* 2015.
- 58. Haley DF, Lucas J, Golin CE, et al. Retention strategies and factors associated with missed visits among low income women at increased risk of HIV acquisition in the US (HPTN 064). *AIDS patient care and STDs* 2014; **28**(4): 206-17.

- 59. Holtzman CW, Shea JA, Glanz K, et al. Mapping patient-identified barriers and facilitators to retention in HIV care and antiretroviral therapy adherence to Andersen's Behavioral Model. *AIDS care* 2015; **27**(7): 817-28.
- 60. Naar-King S, Outlaw A, Green-Jones M, Wright K, Parsons JT. Motivational interviewing by peer outreach workers: a pilot randomized clinical trial to retain adolescents and young adults in HIV care. *AIDS care* 2009; **21**(7): 868-73.
- 61. Nelsen A, Gupta S, Trautner BW, et al. Intention to adhere to HIV treatment: a patient-centred predictor of antiretroviral adherence. *HIV medicine* 2013; **14**(8): 472-80.
- 62. Remien RH, Stirratt MJ, Dolezal C, et al. Couple-focused support to improve HIV medication adherence: a randomized controlled trial. *AIDS* 2005; **19**(8): 807-14.
- 63. Centers for Disease Control and Prevention. Comprehensive Risk Counseling and Services for Persons Living with HIV. 2012. https://effectiveinterventions.cdc.gov/docs/default-source/public-health-strategies-docs/CRCS\_4\_PERSONS\_LIVING\_WITH\_HIV\_Procedur al Guide 8-09 sflb Updated 12-927.pdf?sfvrsn=0 (accessed August 26 2014).
- 64. Gelberg L, Andersen RM, Leake BD. The Behavioral Model for Vulnerable Populations: application to medical care use and outcomes for homeless people. *Health services research* 2000; **34**(6): 1273-302.
- 65. Stein JA, Andersen R, Gelberg L. Applying the Gelberg-Andersen behavioral model for vulnerable populations to health services utilization in homeless women. *Journal of health psychology* 2007; **12**(5): 791-804.
- 66. Remien RH, Stirratt MJ, Dognin J, Day E, El-Bassel N, Warne P. Moving from theory to research to practice. Implementing an effective dyadic intervention to improve antiretroviral adherence for clinic patients. *J Acquir Immune Defic Syndr* 2006; **43 Suppl 1**: S69-78.
- 67. Robbins RN, Mellins CA, Leu CS, et al. Enhancing Lay Counselor Capacity to Improve Patient Outcomes with Multimedia Technology. *AIDS and behavior* 2015.
- 68. Berry M, Raymond HF, Kellogg T, McFarland W. The Internet, HIV serosorting and transmission risk among men who have sex with men, San Francisco. *AIDS* 2008; **22**(6): 787-9.
- 69. Berry M, Raymond HF, McFarland W. Same race and older partner selection may explain higher HIV prevalence among black men who have sex with men. *AIDS* 2007; **21**(17): 2349-50.
- 70. Ma X, Zhang Q, He X, et al. Trends in prevalence of HIV, syphilis, hepatitis C, hepatitis B, and sexual risk behavior among men who have sex with men. Results of 3 consecutive respondent-driven sampling surveys in Beijing, 2004 through 2006. *J Acquir Immune Defic Syndr* 2007; **45**(5): 581-7.
- 71. Raymond HF, Kajubi P, Kamya MR, Rutherford GW, Mandel JS, McFarland W. Correlates of unprotected receptive anal intercourse among gay and bisexual men: Kampala, Uganda. *AIDS and behavior* 2009; **13**(4): 677-81.
- 72. Herek GM, Cogan JC, Gillis JR, Glunt EK. Correlates of internalized homophobia in a community sample of lesbians and gay men. *Journal of the Gay and Lesbian Medical Association* 1997; **2**: 17–25.


- 73. Pence BW, Gaynes BN, Whetten K, Eron JJ, Jr., Ryder RW, Miller WC. Validation of a brief screening instrument for substance abuse and mental illness in HIV-positive patients. *J Acquir Immune Defic Syndr* 2005; **40**(4): 434-44.
- 74. Whetten K, Reif S, Swartz M, et al. A brief mental health and substance abuse screener for persons with HIV. *AIDS patient care and STDs* 2005; **19**(2): 89-99.
- 75. Wilson IB, Fowler FJ, Jr., Cosenza CA, et al. Cognitive and field testing of a new set of medication adherence self-report items for HIV care. *AIDS and behavior* 2014; **18**(12): 2349-58.
- 76. Heckathorn D. Respondent-Driven Sampling II: Deriving Valid Population Estimates from Chain-Referral Samples of Hidden Populations. *Social Problems* 2002; **49**(1): 11-34.
- 77. Garnett GP, Cousens S, Hallett TB, Steketee R, Walker N. Mathematical models in the evaluation of health programmes. *Lancet* 2011; **378**(9790): 515-25.
- 78. Boily MC, Masse B, Alsallaq R, et al. HIV treatment as prevention: considerations in the design, conduct, and analysis of cluster randomized controlled trials of combination HIV prevention. *PLoS medicine* 2012; **9**(7): e1001250.
- 79. Alam SJ, Romero-Severson E, Kim JH, Emond G, Koopman JS. Dynamic sex roles among men who have sex with men and transmissions from primary HIV infection. *Epidemiology* 2010; **21**(5): 669-75.
- 80. Goodreau SM, Goicochea LP, Sanchez J. Sexual role and transmission of HIV Type 1 among men who have sex with men, in Peru. *The Journal of infectious diseases* 2005; **191** Suppl 1: S147-58.
- 81. Sullivan PS, Carballo-Dieguez A, Coates T, et al. Successes and challenges of HIV prevention in men who have sex with men. *Lancet* 2012; **380**(9839): 388-99.
- 82. Cassels S, Menza TW, Goodreau SM, Golden MR. HIV serosorting as a harm reduction strategy: evidence from Seattle, Washington. *AIDS* 2009; **23**(18): 2497-506.
- 83. Wilson DP, Regan DG, Heymer KJ, Jin F, Prestage GP, Grulich AE. Serosorting may increase the risk of HIV acquisition among men who have sex with men. *Sexually transmitted diseases* 2010; **37**(1): 13-7.
- 84. Rosenberg ES, Millett GA, Sullivan PS, Del Rio C, Curran JW. Understanding the HIV disparities between black and white men who have sex with men in the USA using the HIV care continuum: a modeling study. *The lancet HIV* 2014; **1**(3): e112-e8.
- 85. Koppenhaver RT, Sorensen SW, Farnham PG, Sansom SL. The cost-effectiveness of preexposure prophylaxis in men who have sex with men in the United States: an epidemic model. *J Acquir Immune Defic Syndr* 2011; **58**(2): e51-2.
- 86. Gomez GB, Borquez A, Caceres CF, et al. The potential impact of pre-exposure prophylaxis for HIV prevention among men who have sex with men and transwomen in Lima, Peru: a mathematical modelling study. *PLoS medicine* 2012; **9**(10): e1001323.
- 87. Gray RT, Prestage GP, Down I, et al. Increased HIV testing will modestly reduce HIV incidence among gay men in NSW and would be acceptable if HIV testing becomes convenient. *PloS one* 2013; **8**(2): e55449.
- 88. Khanna AS, Goodreau SM, Gorbach PM, Daar E, Little SJ. Modeling the impact of post-diagnosis behavior change on HIV prevalence in Southern California men who have sex with men (MSM). *AIDS and behavior* 2014; **18**(8): 1523-31.

- 89. Kato M, Granich R, Bui DD, et al. The potential impact of expanding antiretroviral therapy and combination prevention in Vietnam: towards elimination of HIV transmission. *J Acquir Immune Defic Syndr* 2013; **63**(5): e142-9.
- 90. Sood N, Wagner Z, Jaycocks A, Drabo E, Vardavas R. Test-and-treat in Los Angeles: a mathematical model of the effects of test-and-treat for the population of men who have sex with men in Los Angeles County. *Clinical infectious diseases : an official publication of the Infectious Diseases Society of America* 2013; **56**(12): 1789-96.
- 91. Granich RM, Gilks CF, Dye C, De Cock KM, Williams BG. Universal voluntary HIV testing with immediate antiretroviral therapy as a strategy for elimination of HIV transmission: a mathematical model. *Lancet* 2009; **373**(9657): 48-57.
- 92. Goodreau SM, Carnegie NB, Vittinghoff E, et al. What drives the US and Peruvian HIV epidemics in men who have sex with men (MSM)? *PloS one* 2012; 7(11): e50522.
- 93. Turner KM, Garnett GP, Ghani AC, Sterne JA, Low N. Investigating ethnic inequalities in the incidence of sexually transmitted infections: mathematical modelling study. *Sexually transmitted infections* 2004; **80**(5): 379-85.
- 94. Mitchell KM, Foss AM, Prudden HJ, et al. Who mixes with whom among men who have sex with men? Implications for modelling the HIV epidemic in southern India. *Journal of theoretical biology* 2014; **355**: 140-50.
- 95. Eaton JW, Hallett TB. Why the proportion of transmission during early-stage HIV infection does not predict the long-term impact of treatment on HIV incidence. *Proceedings of the National Academy of Sciences of the United States of America* 2014; **111**(45): 16202-7.
- 96. Lodi S, Phillips A, Touloumi G, et al. Time from human immunodeficiency virus seroconversion to reaching CD4+ cell count thresholds <200, <350, and <500 Cells/mm(3): assessment of need following changes in treatment guidelines. *Clinical infectious diseases : an official publication of the Infectious Diseases Society of America* 2011; **53**(8): 817-25.
- 97. Baggaley RF, White RG, Boily MC. HIV transmission risk through anal intercourse: systematic review, meta-analysis and implications for HIV prevention. *International journal of epidemiology* 2010; **39**(4): 1048-63.
- 98. Boily MC, Baggaley RF, Wang L, et al. Heterosexual risk of HIV-1 infection per sexual act: systematic review and meta-analysis of observational studies. *The Lancet Infectious diseases* 2009; **9**(2): 118-29.
- 99. Jin F, Jansson J, Law M, et al. Per-contact probability of HIV transmission in homosexual men in Sydney in the era of HAART. *AIDS* 2010; **24**(6): 907-13.
- 100. Fideli US, Allen SA, Musonda R, et al. Virologic and immunologic determinants of heterosexual transmission of human immunodeficiency virus type 1 in Africa. *AIDS research and human retroviruses* 2001; **17**(10): 901-10.
- 101. Jean K, Gabillard D, Moh R, et al. Effect of early antiretroviral therapy on sexual behaviors and HIV-1 transmission risk among adults with diverse heterosexual partnership statuses in Cote d'Ivoire. *The Journal of infectious diseases* 2014; **209**(3): 431-40.
- 102. Quinn TC, Wawer MJ, Sewankambo N, et al. Viral load and heterosexual transmission of human immunodeficiency virus type 1. Rakai Project Study Group. *The New England journal of medicine* 2000; **342**(13): 921-9.

- 103. Mills E, Cooper C, Anema A, Guyatt G. Male circumcision for the prevention of heterosexually acquired HIV infection: a meta-analysis of randomized trials involving 11,050 men. *HIV medicine* 2008; **9**(6): 332-5.
- 104. Hughes JP, Baeten JM, Lingappa JR, et al. Determinants of per-coital-act HIV-1 infectivity among African HIV-1-serodiscordant couples. *The Journal of infectious diseases* 2012; **205**(3): 358-65.
- 105. Weller S, Davis K. Condom effectiveness in reducing heterosexual HIV transmission. *The Cochrane database of systematic reviews* 2002; (1): CD003255.
- 106. Poole D, Raftery AE. Inference for Deterministic Simulation Models: The Bayesian Melding Approach. *Journal of the American Statistical Association* 2000; **95**: 1244-55.
- 107. Hallett TB, Gregson S, Mugurungi O, Gonese E, Garnett GP. Assessing evidence for behaviour change affecting the course of HIV epidemics: a new mathematical modelling approach and application to data from Zimbabwe. *Epidemics* 2009; **1**(2): 108-17.
- 108. Pickles M, Boily MC, Vickerman P, et al. Assessment of the population-level effectiveness of the Avahan HIV-prevention programme in South India: a preplanned, causal-pathway-based modelling analysis. *The Lancet Global health* 2013; **1**(5): e289-99.
- 109. Vickerman P, Platt L, Hawkes S. Modelling the transmission of HIV and HCV among injecting drug users in Rawalpindi, a low HCV prevalence setting in Pakistan. *Sexually transmitted infections* 2009; **85 Suppl 2**: ii23-30.
- 110. Boily MC, Lowndes CM, Vickerman P, et al. Evaluating large-scale HIV prevention interventions: study design for an integrated mathematical modelling approach. *Sexually transmitted infections* 2007; **83**(7): 582-9.
- 111. Mishra S, Pickles M, Blanchard JF, Moses S, Boily MC. Distinguishing sources of HIV transmission from the distribution of newly acquired HIV infections: why is it important for HIV prevention planning? *Sexually transmitted infections* 2014; **90**(1): 19-25.
- 112. Mishra S, Pickles M, Blanchard JF, Moses S, Shubber Z, Boily MC. Validation of the modes of transmission model as a tool to prioritize HIV prevention targets: a comparative modelling analysis. *PloS one* 2014; **9**(7): e101690.

**APPENDICES** 

APPENDIX I: SCHEDULE OF STUDY VISITS, EVALUATIONS AND PROCEDURES

| | Screening | Enrollment<br>(M0) | Monthly<br>Contact <sup>1</sup> | Follow-up<br>(M3, M6, M9,<br>M12, M18) | Final (M24) |
|---|---|---|---|---|---|
| Administrative and Behavioral Evaluations/Pro | ocedures | | | | |
| Informed consent | X | X | | | |
| Release of medical information | | X | | | |
| Contact/locator information | X | X | I | X | X |
| Questionnaire administration (see Appendix II) | X | X | | | X |
| Recruiter training | X | | | | |
| Coupon reimbursement | X | | | | |
| Social impact assessment | $X^2$ | | I | X | X |
| Pre- and post-test HIV counseling, including HIV/STI risk reduction counseling | X | $X^3$ | | | |
| Offer of partner HIV counseling and testing | | X | | X | X |
| Coupon disbursement | $X^4$ | | | | |
| Case manager (CM) intervention | | I | I | I | I |
| Exit interview | | | | | X |
| Clinical Evaluations/Procedures | | | | | |
| Blood collection | X | X | | X | X |
| Syphilis treatment or referral, if indicated | X | X <sup>5</sup> | | | $X^6$ |
| HCV treatment or referral, if indicated | X | X <sup>5</sup> | | | |
| Laboratory Evaluations/Procedures | • | | | | |
| HIV testing | $X^{7,9}$ | | | | |
| Hepatitis C virus testing | X <sup>7</sup> | | | | |
| Syphilis testing | X8 | | | | X |
| CD4 cell count testing | $X^9$ | | | X | X |
| HIV viral load testing | $X^9$ | | | X | X |
| Plasma storage <sup>10</sup> | | X | | X | X |

Note: Monthly visits will be defined as a predetermined number of weeks, as described in the SSP. In addition, in special cases, the screening and enrollment visits may take place on the same day (see SSP).

Note: At the start of the study, plasma was stored at screening (not at enrollment). If plasma is not available from enrollment, plasma from screening may be used for HPTN LC testing

X, all participants; I, CM intervention arm only.

<sup>&</sup>lt;sup>1</sup>Monthly contact is only provided to participants in the CM intervention arm; these interactions may be conducted in person or by phone, text message or email.

<sup>&</sup>lt;sup>2</sup>Social impact assessments will not be collected until after first study encounter.

<sup>&</sup>lt;sup>3</sup>Test results may be given at the enrollment visit, including post-testing counseling

<sup>&</sup>lt;sup>4</sup>In special cases, participants may receive additional coupons after screening. See SSP for detailed instructions.

<sup>&</sup>lt;sup>5</sup>Treatment or referral for HCV and/or Syphilis treatment may be given at the enrollment visit.

<sup>&</sup>lt;sup>6</sup>If the syphilis test is positive, participants will be given their test results and referred for care via site standards.

<sup>&</sup>lt;sup>7</sup>Procedures for HIV and HCV testing are described in the SSP Manual.

<sup>&</sup>lt;sup>8</sup>Syphilis testing will be performed using blood specimens according to local standards.

<sup>&</sup>lt;sup>9</sup>If HIV positive by self-report, clinic record or by having a reactive HIV rapid test at screening, blood will be collected for HIV confirmatory testing, HIV viral load and CD4+ cell count.

<sup>&</sup>lt;sup>10</sup>Stored plasma will be used for Quality Assurance testing and other assessments at the HPTN LC (see Section 9.2). These assessments will be performed retrospectively; results will not be returned to study sites or participants except as noted in Section 9.2.

# APPENDIX II: SCHEDULE OF OUESTIONNAIRE DOMAIN ADMINISTRATION

| Questionnaire Domain | Screening | Enrollment (M0) (Intervention participants [CM Intervention and SOC control arms]) | Final (M24) (Intervention participants [CM Intervention and SOC control arms]) |
|---|---|---|---|
| Demographics | X | | |
| PrEP/PEP/ART use | X | | |
| HIV testing history | X | | |
| Engagement in LGBT community | X | | |
| Post-recruitment questions* | X | | |
| Health care utilization | X | | X |
| Sexual matrix module / sexual risk behavior | X | | X |
| Stigma | X | | X |
| Substance use and mental health | | X | X |
| Medication adherence | | | X |
| Exit Interview Questionnaire | | | X** |

<sup>\*</sup>These questions will only be asked of those who were given coupons to distribute and who distributed, or attempted to distribute, them. For those enrolled, this questionnaire may be administered at or after enrollment, as applicable.


\

<sup>\*\*</sup>The exit interview will be conducted with both participants and CMs.

APPENDIX III: INFORMED CONSENT TEMPLATES

# **Enhancing Recruitment, Linkage to Care and Treatment for HIV-Infected Men Who Have Sex with Men (MSM) in the United States**

#### **HPTN 078**

Version 2.0 July 3, 2017 DAIDS Document ID: 11995

#### HIV SCREENING INFORMED CONSENT FORM

**Sponsored by:** Division of AIDS (DAIDS), United States (US) National Institute of Allergy and Infectious Diseases (NIAID), US National Institute of Mental Health (NIMH), US National Institute on Drug Abuse (NIDA) and US National Institutes of Health (NIH).

PRINCIPAL INVESTIGATOR: [Insert Name]

**PHONE:** [Insert Number]

**INTRODUCTION:** You are being asked to take part in a research study. This study is looking at the best way to find men who have sex with men (MSM) and transgender women, who may be at risk for getting HIV (Human Immunodeficiency Virus). To find out if you are eligible for this study, a rapid HIV test will be done to test for HIV. [Sites may add reference to the inclusion of transgender women to the extent that they want, may change third person pronouns (eg., he to they) as they see fit for their site or may choose to have a separate consent for transgender women.]

If your rapid test is positive for HIV, repeat testing is needed to confirm (prove) this result. If your second sample is proved to be positive for HIV, it means that you have HIV. This means that you can pass the virus to others by sexual contact, by sharing needles, and by donating blood and organs. A negative rapid test means that you do not have HIV but should be tested again if you have been exposed within the last 3-6 months.

**YOUR PARTICIPATION IS VOLUNTARY:** You may refuse to be screened. You may also refuse the HIV test or to give your contact information. You may withdraw your consent for screening at any time.

**SCREENING PROCESS:** You will receive a rapid HIV test. The rapid test will use a drop of blood from your finger or a swab from the inside of your mouth. You will be provided pre- and post-test counseling [sites to revise per their requirements]. We will also ask for your contact information so that we can reach you when your test results are complete. [Sites to add expected duration]. When your results are ready, you will be scheduled for an appointment. This appointment will be to discuss your results and receive further testing, if you choose.

If you already know that you are HIV positive, you don't need to take a rapid HIV test. If you would like, you may still give your contact information to be scheduled for an appointment. This appointment will do further screening to see if you are eligible for this study.

**RISKS AND/OR DISCOMFORTS**: You may be nervous while you are waiting for your HIV test result. If the test shows that you have HIV, you may worry about your health and future. You will receive counseling before and after the test to help address your concerns [sites to revise per their requirements].

We will make every effort to protect the privacy of your HIV test results. However, it is possible that others may learn that you are part of this screening. They may think that you are infected with HIV. Because of this you could have trouble finding or keeping a job. You could also have problems with your family, friends and community.

There is also a small risk of infection if you have the finger stick for blood draw.

**BENEFITS:** The benefits of being screened for HIV include knowing your HIV status. Finding HIV infection early can also be important for your treatment.

**ALTERNATIVES TO PARTICIPATION:** [Sites to include/alter the following if applicable: If you would like, we will tell you how to get HIV testing anonymously at other places.]

**REIMBURSEMENT:** You will receive [site to add amount] for your time to be tested for HIV today. [Sites to insert information about local reimbursement for the study.]

**CONFIDENTIALITY:** All of your contact information will be kept private. Your test results will also be kept private. This information will not be shared with others. All records will be stored in locked files at the study clinic.

[Sites to include/amend the following if applicable:] [Local/state/national] regulations require study staff to report the names of people who test positive for HIV to the [local health authority]. Outreach workers from the [health authority] may then contact you about telling your partners, since they also should be tested. If you do not want to tell your partners yourself, the outreach workers will contact them, according to the privacy guidelines of the [health authority].

**PROBLEMS OR QUESTIONS:** If you ever have any questions about the screening procedures, or if you have a research-related injury, you should contact [insert name of the investigator or other study staff] at [insert telephone number and/or physical address].

If you have questions about your rights as a research participant, you should contact [insert name or title of person on the IRB or other organization appropriate for the site] at [insert physical address and telephone number].

If you have read this consent form, or had it read and explained to you, and you understand the information, and you voluntarily agree to test for HIV and give your contact information, please sign your name or make your mark below.

| Participant Name (print) | Participant Signature and Date [sites to include if applicable] consent or assert |
|---|---|
| Study Staff Conducting Consent Discussion (print) | Study Staff Signature and Date |
| Witness Name (print) (As appropriate) | Witness Signature and Date |

# Enhancing Recruitment, Linkage to Care and Treatment for HIV-Infected Men Who Have Sex with Men (MSM) in the United States

#### **HPTN 078**


#### SCREENING INFORMED CONSENT FORM

**Sponsored by:** Division of AIDS (DAIDS), United States (US) National Institute of Allergy and Infectious Diseases (NIAID), US National Institute of Mental Health (NIMH), US National Institute on Drug Abuse (NIDA) and US National Institutes of Health (NIH).

PRINCIPAL INVESTIGATOR: [Insert Name]

**PHONE:** [Insert Number]

#### INTRODUCTION

You are being asked to take part in a research study. This study is designed to find the best way to find men who have sex with men (MSM) and offer them HIV testing. Joining this study is voluntary. You may refuse to join, or you may withdraw your consent to be in the study, for any reason. This study is for MSM and transgender women, who may be at risk for getting Human Immunodeficiency Virus, or HIV. HIV is the virus that causes Acquired Immunodeficiency Syndrome, or AIDS. [Sites may add reference to the inclusion of transgender women to the extent that they want, may change third person pronouns (eg., he to they) as they see fit for their site or may choose to have a separate consent for transgender women.]

Before you decide whether to join the study, we would like to explain the purpose of the screening, the risks and benefits, and what is expected of you.

#### YOUR PARTICIPATION IS VOLUNTARY

This consent form gives information about the screening. Once you understand the screening, and if you agree to take part, you will be asked to sign your name or make your mark on this form. You will be offered a copy of this form to keep.

Before you learn about screening, it is important that you know the following:

- Your participation is voluntary. You do not have to take part in any of the screening tests, questionnaires or procedures.
- You may decide not to take part in screening, or you may decide to leave the screening at any time.
- If you decide not to take part in the screening, you can still join another study at a later time if there is one available and you qualify.
- If you decide not to take part in the screening, or decide to stop participating at any time, there will be no penalty or loss of the normal benefits provided to you at our clinic.

## PURPOSE OF THE SCREENING

The purpose of the screening is to find MSM using a method called "respondent driven sampling" or "RDS." In RDS, we ask MSM to invite other MSM they know to come to our clinic for screening. We will also invite MSM to take part in this study that we find in other ways.

We plan to screen about 2700 people from four US cities (about 675 in each participating city) in two years. During screening, we will test MSM for HIV, hepatitis C virus and syphilis. We will also ask each MSM to complete a questionnaire. If we find MSM who are HIV-infected, we may invite them to take part in another study. This other study is testing whether case manager support can help MSM receive regular HIV care and regularly take their HIV medication.

Information from the screening procedures will be used to prevent the spread of HIV in the MSM community.

#### SCREENING PROCEDURES

If you agree to participate, you will be asked to take part in up to three screening visits.

Screening will happen after you read, discuss, understand, and sign this form. We will help you understand the form and answer your questions before you sign this form. The procedures done during Screening will take about [sites to fill in the amount of time] hours each time.

#### During screening:

- We will confirm where you live and how to contact you.
- We will ask you to answer a questionnaire. This questionnaire will ask you about yourself (like your age and race) and your sexual behavior and partners. It will also ask you about your use of HIV drugs, HIV testing history and health care use. Finally, it will ask you about your involvement in the lesbian, gay, bisexual and transgender (LGBT) community and stigma you may have faced because you are an MSM.
- We will ask you if you have had any problems because you are a part of this screening.
- We will talk to you about HIV and other infections that can be spread sexually. We will give you information to help you protect yourself from getting them or passing them on to others.
- We may give you a rapid HIV test. The rapid test will use a drop of blood from your finger or arm or a swab from the inside of your mouth. If your rapid test is positive for HIV, repeat testing is needed to confirm (prove) this result. If your second sample is proved to be positive for HIV, it means that you have HIV. A negative rapid test means that you do not have HIV but should be tested again if you have been exposed within the last 3-6 months.
- We will collect a small amount of blood about 33 mL = about 6 teaspoons) to test for hepatitis C virus (HCV) and syphilis.
- If you are HIV-infected, a small amount of blood (about 14 mL = about 3 teaspoons) will be collected to make sure you have HIV. This blood will also be used to measure your CD4 cell count and viral load. These tests tell us how much HIV is in your blood (viral load) and how much the virus has affected your ability to fight the virus (CD4).
- We may give you coupons and ask you to invite MSM you know to come to the clinic for screening.

- We will give you the results of your HIV, hepatitis C virus and syphilis tests. If you have any of these infections, you will be referred for treatment [sites to add specifics about how this will take place at their site].
- If we can't tell if you are infected or not after your HIV tests, you will be referred for further testing and care.
- If you were asked to invite people you know to come for HIV testing, we will ask you questions about who you invited.

**If you are HIV-uninfected:** If your HIV test results show that you aren't infected, we will give you information about how to prevent getting HIV.

If you are HIV-infected: If your HIV test results show that you are infected, we will check your viral load test to see if you are eligible for another study. If so, we may ask you if you are interested in being in the study. The study is testing if case manager support can help those who are HIV-infected. If you do not want to take part in this study, we will tell you where you can go to receive HIV care.

#### RISKS AND/OR DISCOMFORTS

#### **Blood Draws**

Taking blood samples may cause some pain, bruise your arm, or make you feel lightheaded. In rare cases, you may faint. There is also a small chance of infection when blood is drawn.

## **HIV Testing and Potential Social Harm**

You may be nervous while you are waiting for your HIV test result. If the tests show that you have HIV, you may worry about your health and future. You will receive counseling before and after the test to help address your concerns. We will make every effort to protect your confidentiality during the study. However, it is possible that others may learn that you are part of this screening. They may think that you are infected with HIV or are at high risk for infection with HIV. Because of this you could have trouble finding or keeping a job. You could also have problems with your family, friends and community.

#### **Sensitive Questions**

The questions we will ask you about your sexual behavior and partners or about stigma you may have faced may make you feel uneasy. However, you do not have to answer any question that you do not want to. You can also stop answering the questions at any time.

# **BENEFITS**

We will test you for HIV, hepatitis C virus and syphilis. If you have any of these infections, we will help you receive care and treatment. We will also tell you how to avoid passing them on to your sexual partners. The counseling you get during this study may help you avoid HIV and other infections that can be spread sexually.

You may not receive any other direct benefit from being in this study. You or others in your community may benefit from these screening activities in the future. The information found during screening may help prevent HIV and other infections in the MSM community.
## **NEW INFORMATION**

You will be told about any new information that might affect your willingness to take part in screening. You will also be told when the results of the study may be ready, and how to learn about them.

## WHY YOU MAY BE WITHDRAWN FROM SCREENING WITHOUT YOUR CONSENT

You may be withdrawn from screening without your consent if any of the following occur:

- You are unable or unwilling to follow all of the screening procedures or instructions.
- Screening is stopped or canceled.
- The study staff feels that taking part in the screening activities would be harmful to you.
- You are not able to attend the screening visits or complete all of the screening procedures.
- Other reasons, as decided by the study staff.

#### ALTERNATIVES TO PARTICIPATION

You may choose not to participate in the study. [Sites to include/amend the following if applicable: You do not need to participate in the screening activities to be tested for HIV at our site. If you wish, we will tell you how to get HIV counseling and testing at other places.]

#### **COSTS TO YOU**

There will be no cost to you for any screening visits, laboratory tests or other procedures.

#### REIMBURSEMENT

You will receive [site to add amount] for your time, effort, and travel to and from the clinic for each scheduled screening visit. [Sites to insert information about local reimbursement for the study.]

## CONFIDENTIALITY

All the information you give us as part of this study will be kept private. All your laboratory test results will also be kept private. You will get a unique study identification number that will be used instead of your name on your documents. However, at every screening visit we will ask you to identify yourself. This is to make sure that it is you who provides samples and information to us. Also, we want to make sure that no other person than you can get your confidential laboratory test results. Only the study staff will be able to see records that identify you by name. This information will not be shared with others. All records will be stored in locked files at the study clinic. Results of your laboratory tests will be made available only to you when you visit the clinic. Your name will never be used in any publication or presentation about these screening activities.

[Sites to modify this suggested language as appropriate:] If you are under 18 years old, we [must/do not need to] inform your parents or guardian about the results of your HIV and syphilis tests, unless you would like us to tell them. If you are under 18 years old, we [must/do not need to] inform your parents or guardian about the results of your hepatitis C (HCV) test, unless you would like us to tell them. If [we must / you choose to have us] inform them of these test results, we will talk to you about the best way to inform them before we do so.

Your records may be looked at by the sponsor of the study, the US National Institutes of Health (NIH). They may also be looked at by NIH representatives, other government and regulatory authorities, [insert name of site] IRB/EC, study staff, study monitors and [insert applicable local regulatory authorities].

In addition to the efforts made by the study staff to help keep your personal information confidential, we have obtained a Certificate of Confidentiality from the U.S. Federal Government. This Certificate protects researchers from being forced to tell people who are not connected with this study, such as the court system, about your participation. The Certificate of Confidentiality does not prevent you from releasing information about yourself and your participation in the study. The Certificate cannot be used to resist a demand for information from personnel of the US Government that is used for auditing or evaluation of federally funded projects or for information that must be disclosed in order to meet the requirements of the US FDA. Even with the Certificate of Confidentiality, if the study staff learns of possible child abuse and/or neglect or a risk of harm to you or others, we will tell the proper authorities.

A description of this study will be on <a href="www.ClinicalTrials.gov">www.ClinicalTrials.gov</a>. This web site will not include information that can identify you. At most, the web site will include a summary of the results. You can search this web site at any time.

[Sites to include/amend the following if applicable:] In this study, you will be tested for HIV, hepatitis C virus and syphilis. [Local/state/national] regulations require study staff to report the names of people who test positive for [HIV and other infections [sites should add that HCV and syphilis are reportable diseases if this is true for their location] to the [local health authority]. Outreach workers from the [health authority] may then contact you about telling your partners, since they also should be tested. If you do not want to tell your partners yourself, the outreach workers will contact them, according to the privacy guidelines of the [health authority].

## RESEARCH-RELATED INJURY

[Sites to specify institutional policy:] It is unlikely that you will be injured because of your study participation. If you are injured, the [institution] will give you immediate necessary treatment for your injuries. You [will/will not] have to pay for this treatment. You will be told where you can get further treatment for your injuries. There is no program to pay money or give other forms of payment for such injuries either through this institution or the US NIH. You do not give up any legal rights by signing this consent form.

## PROBLEMS OR OUESTIONS

If you ever have any questions about the screening activities, or if you have a research-related injury, you should contact [insert name of the investigator or other study staff] at [insert telephone number and/or physical address].

If you have questions about your rights as a research participant, you should contact [insert name or title of person on the IRB or other organization appropriate for the site] at [insert physical address and telephone number].

# **SIGNATURE PAGE**

Enhancing Recruitment, Linkage to Care and Treatment for HIV-Infected Men Who Have Sex with Men (MSM) in the United States

## **HPTN 078**


# SCREENING INFORMED CONSENT FORM

If you have read this consent form, or had it read and explained to you, and you understand the information, and you voluntarily agree to complete the screening activities, please sign your name or make your mark below.

| Participant Name (print) | Participant Signature and Date [sites to include if applicable] consent or assen |
|---|---|
| Study Staff Conducting Consent Discussion (print) | Study Staff Signature and Date |
| Witness Name (print) (As appropriate) | Witness Signature and Date |

# Enhancing Recruitment, Linkage to Care and Treatment for HIV-Infected Men Who Have Sex with Men (MSM) in the United States

# **HPTN 078**


## ENROLLMENT INFORMED CONSENT FORM

**Sponsored by:** Division of AIDS (DAIDS), United States (US) National Institute of Allergy and Infectious Diseases (NIAID), US National Institute of Mental Health (NIMH), US National Institute on Drug Abuse (NIDA) and US National Institutes of Health (NIH).

PRINCIPAL INVESTIGATOR: [Insert Name]

**PHONE:** [Insert Number]

#### INTRODUCTION

You are being asked to take part in a research study. This study is testing if support from a case manager can help HIV-infected people receive regular HIV care and regularly take their HIV medication. Joining this study is voluntary. You may refuse to join, or you may withdraw your consent to be in the study, for any reason. This research study is for men who have sex with men (MSM) and transgender women, who have <u>Human Immunodeficiency Virus</u>, or HIV. HIV is the virus that causes <u>Acquired Immunodeficiency Syndrome</u>, or AIDS. [Sites may add reference to the inclusion of transgender women to the extent that they want, may change third person pronouns (eg., he to they) as they see fit for their site or may choose to have a separate consent for transgender women.]

Before you decide whether to join the study, we would like to explain the purpose of the study, the risks and benefits, and what is expected of you.

## YOUR PARTICIPATION IS VOLUNTARY

This consent form gives information about the study you are being invited to join. Once you understand the study, and if you agree to take part, you will be asked to sign your name or make your mark on this form. You will be offered a copy of this form to keep.

Before you learn about the study, it is important that you know the following:

- Your participation is voluntary. You do not have to take part in any of the tests, questionnaires or procedures in the study.
- You may decide not to take part in the study, or you may decide to leave the study at any time.
- If you decide not to take part in the study, you can still join another study at a later time if there is one available and you qualify.
- If you decide not to take part in the study, or decide to stop participating at any time, there will be no penalty or loss of the normal benefits provided to you at our clinic.

# PURPOSE OF THE STUDY

The purpose of this study is to find out if support from a case manager can help HIV-infected people receive regular HIV care and regularly take their HIV medication.

The purpose of this study is also to help researchers understand how HIV spreads in the community. We will look at the different types of virus found in the blood samples of different people in the community who are living with HIV. In science, we call this phylogenetics.

#### STUDY GROUPS

We plan to enroll 356 HIV-infected men and follow them for two years. Half of the participants will receive the intervention (support from a case manager [CM]) and the other half will not. At the end of the study, the two groups will be compared to see if the CM support helped participants stay in HIV care and take their HIV drugs regularly.

You will be "randomized" to either the group who will get case manager support or the group who will get the same care that patients normally get to stay in HIV care and take their HIV drugs regularly. "Randomization" means that you are put into a group by chance. It is like flipping a coin. You have will an equal chance of being in either group. Both groups are important to the study.

# **CM Intervention Group**

If you are in the CM <u>intervention group</u>, you will receive support from a case manager who will help you link to and stay in HIV care. When you are ready, the case manager will also help you start HIV medication and take it properly. The help from the case manager will be specific to your needs.

# Standard-of-Care (SOC) Control Group

If you are in the SOC <u>control group</u>, you will get the same care that patients normally get to stay in HIV care and take their HIV drugs properly.

#### **Co-Enrollment in Other Studies**

While you are in this study, you may not take part in other studies that help you link to HIV care or take your HIV medication properly.

## STUDY PROCEDURES

If you join the study, you will be asked to take part in 7 study visits over two years. If you are in the case manager group, you will also be contacted about the study monthly.

#### **Enrollment Visit**

Your enrollment visit will happen after you read, understand, and sign this form. We will help you understand the form and answer your questions before you sign this form. The procedures done at the Enrollment Visit will take about [sites to fill in the amount of time] hours.

# During this visit:

• We will confirm where you live and how to contact you.

- We will give you the results of your HIV, hepatitis C virus and syphilis tests if you did not receive them at screening. If you have any of these infections, you will be referred for treatment [sites to add specifics about how this will take place at their site].
- We will ask you to give us permission to review your medical records.
- We will ask you to answer a questionnaire. This questionnaire will ask you about your use of recreational drugs and alcohol. It will also ask about your mental health.
- We will invite you to bring your sexual partner(s) for HIV testing. [Note: Partner testing is conducted outside of the study and results are not recorded.]
- If you are in the case manager group, the study case manager (CM) will talk to you about HIV. They will give you information to help you decide where you would like to go for HIV care and when to start HIV drugs. You will choose how much support you need from the case manager. You can talk with the case-manager by text, email, phone, or in-person. The session with the case manager will be audio-recorded.
- We will collect a small amount of blood (about 34 mL = about 7 teaspoons) which will be stored. This blood will be used to check the results of tests performed at the study site and other study testing. This testing will give us information about the HIV virus and how the virus spreads in the community. The blood may also be used to test for the presence of HIV drugs and to learn more about how the body responds to HIV infection. If you have hepatitis C, the blood may also be used for testing to learn more about the hepatitis C virus and how it spreads in the community. Results from testing using stored samples will not be returned to you or the study site.

# **Monthly Contact**

If you are in the case manager group, you will be contacted every month to confirm where you live and how to find you. We will ask if you are having any problems with your health or your HIV medication. We will ask you if you have had any problems because you are a part of this study. You may choose to have us call, email or text you every month. You can also ask to meet with the case manager monthly, or more often, if you want more support.

# **Follow-up Visits**

You will be asked to return to the clinic for a total of 5 Follow-up Visits. The procedures done at the Follow-up Visits will take about [sites to fill in the amount of time] hours.

# During this visit:

- We will confirm where you live and how to contact you.
- We will ask you if you have had any problems because you are a part of this study.
- We will invite you to bring your sexual partner(s) for HIV testing.
- We will collect a small amount of blood (about 34 mL = about 7 teaspoons) to do CD4 cell count and viral load testing. Some of the blood will be stored for additional testing. These tests will give us information about the HIV virus and how the virus spreads in the community. The blood may also be used to test for the presence of HIV drugs and to learn more about how the body responds to HIV infection. If you have hepatitis C, the blood may also be used for testing to learn more about the hepatitis C virus and how it spreads in the

community. Results from testing using stored samples will not be returned to you or the study site.

• If you are in the case-manager group, you will meet with the case manager to talk about your HIV care. You will also talk about your HIV medication if you have started taking it. The case manager will help you with any problems you are having. The session with the case manager will be audio-recorded.

#### Final Visit

At the end of two years, you will be asked to return to the clinic for a Final Visit. The procedures done at the Final Visit will take about *[sites to fill in the amount of time]* hours.

# During this visit:

- We will confirm where you live and how to contact you.
- We will ask you to answer a questionnaire. This questionnaire will ask you about your sexual behavior and partners, medication adherence, health care use. It will also ask you about your use of recreational drugs and alcohol, your mental health and stigma you may have faced because you are an MSM.
- We will ask you if you have had any problems because you are a part of this study.
- We will invite you to bring your sexual partner(s) for HIV testing.
- We will ask you to take part in an exit interview. This interview may also include a questionnaire. Both the questionnaire and the interview will ask you about how you felt about being in the study.
- We will collect a small amount of blood (about 40 mL = about 8 teaspoons) to do CD4 cell count, HIV viral load and syphilis testing. Some of this blood will be stored for additional testing. These tests will give us information about the HIV virus and how the virus spreads in the community. The blood may also be used to test for the presence of HIV drugs and to learn more about how the body responds to HIV infection. If you have hepatitis C, the blood may also be used for testing to learn more about the hepatitis C virus and how it spreads in the community. Results from testing using stored samples will not be returned to you or the study site.
- We will contact you when the results of your syphilis test are available. You will be given your results [sites to input information according to site standards]. If your test is positive, you will be referred for care and treatment [sites to input information on site standards].
- If you are in the case-manager group, you will meet with the case manager to talk about your HIV care. You will also talk about your HIV medication if you have started taking it. The case manager will help you with any problems you are having. The session with the case manager will be audio-recorded.

# If You Decide to Leave the Study Early

If you decide to leave the study early (before completing the final study visit), you will be asked to complete a final evaluation. This will include all of the procedures listed for the final visit.

# When You Decide to Start HIV Drugs

If you decide to start taking HIV medication, we will ask your doctors for information about when you started these drugs. We will also ask what your CD4 cell count and HIV viral load test results were at that time.

## **HIV Test Results for Your Sexual Partner**

**If your sexual partner is HIV-uninfected:** If your sexual partner is found to be HIV negative at any study visit, we will give both of you information about how to prevent the spread of HIV.

**If your sexual partner is HIV-infected:** If your sexual partner is found to be HIV positive at any study visit, we will talk to him about what this test result means and where they can receive HIV care.

#### RISKS AND/OR DISCOMFORTS

## **Blood Draws**

Taking blood samples may cause some pain, bruise your arm, or make you feel lightheaded. In rare cases you may faint. There is also a small chance of infection when blood is drawn.

# **Sensitive Questions**

The questions we will ask you about your sexual behavior and partners, recreational drug and alcohol use, your mental health or about stigma you may have faced may make you feel uneasy. However, you do not have to answer any question that you do not want to. You can also stop answering the questions at any time.

# **Potential Social Harm**

We will make every effort to protect your privacy during the study. However, it is possible that others may learn that you are part of the study. They may think that you are infected with HIV. Because of this you could have trouble finding or keeping a job. You could also have problems with your family, friends and community.

# **BENEFITS**

The counseling you get during this study may help you avoid spreading HIV to anyone else. We will offer to test your sexual partner for HIV. We will test you for syphilis. If you have syphilis, we will refer you for care and treatment.

If you are in the CM intervention group, you will receive help from a case manager to stay in HIV care and take your HIV drugs properly.

You may not receive any other direct benefit from being in this study. You or others in your community may benefit from this study in the future. The information found during this study may help prevent HIV and other infections in the MSM community.

#### **NEW INFORMATION**

You will be told about any new information learned during this study that might affect your willingness to take part in the study. You will also be told when the results of the study may be ready, and how to learn about them.

# WHY YOU MAY BE WITHDRAWN FROM THE STUDY WITHOUT YOUR CONSENT

You may be withdrawn from the study without your consent if any of the following occur:

- You are unable or unwilling to follow all of the study procedures or instructions.
- The study is stopped or canceled.
- The study staff feels that staying in the study would be harmful to you.
- You are not able to attend clinic visits or complete all of the study procedures.
- Other reasons, as decided by the study staff.

# ALTERNATIVES TO PARTICIPATION

You may choose not to take part in the study. [Sites to include/amend the following if applicable: There may be other studies going on here or in the community that you may be eligible for. Some of these studies may be able to help you stay in HIV care or take your HIV medication. If you wish, we will tell you about other studies that we know about.]

## **COSTS TO YOU**

There will be no cost to you for any study-related visits, laboratory tests or other procedures.

#### REIMBURSEMENT

You will receive [site to add amount] for your time, effort, and travel to and from the clinic for each scheduled visit. [Sites to insert information about local reimbursement for the study.]

#### CONFIDENTIALITY

All the information you give us as part of this study will be kept private. All your laboratory test results will also be kept private. You will get a unique study identification number that will be used instead of your name on your documents. However, at every study visit we will ask you to identify yourself. This is to make sure that it is you who provides samples and information to us. Also we want to make sure that no other person than you can get your confidential laboratory test results. Only the study staff will be able to see records that identify you by name. This information will not be shared with others. All records will be stored in locked files at the study clinic. Results of your laboratory tests will be made available only to you when you visit the clinic. Your name will never be used in any publication or presentation about the study.

[Sites to modify this suggested language as appropriate:] If you are under 18 years old, we [must/do not need to] inform your parents or guardian about the results of your HIV and syphilis test, unless you would like us to tell them. If you are under 18 years old, we [must/do not need to] inform your parents or guardian about the results of your hepatitis C (HCV) test, unless you would like us to tell them. If [we must / you choose to have us] inform them of these test results, we will talk to you about the best way to inform them before we do so.

Your records may be reviewed by the sponsor of the study, the US National Institutes of Health (NIH). They may also be looked at by NIH representatives, other government and regulatory authorities, [insert name of site] IRB/EC, study staff, study monitors and [insert applicable local regulatory authorities].

In addition to the efforts made by the study staff to help keep your personal information confidential, we have obtained a Certificate of Confidentiality from the U.S. Federal Government.

This Certificate protects researchers from being forced to tell people who are not connected with this study, such as the court system, about your participation. The Certificate of Confidentiality does not prevent you from releasing information about yourself and your participation in the study. The Certificate cannot be used to resist a demand for information from personnel of the US Government that is used for auditing or evaluation of federally funded projects or for information that must be disclosed in order to meet the requirements of the US FDA. Even with the Certificate of Confidentiality, if the study staff learns of possible child abuse and/or neglect or a risk of harm to you or others, we will tell the proper authorities.

A description of this study will be on <u>www.ClinicalTrials.gov</u>. This web site will not include information that can identify you. At most, the web site will include a summary of the results. You can search this web site at any time.

[Sites to include/amend the following if applicable:] In this study, you will be tested for syphilis and your sexual partner may be tested for HIV. [Local/state/national] regulations require study staff to report the names of people who test positive for [HIV and other infections] to the [local health authority]. Outreach workers from the [health authority] may then contact you about telling your partners, since they also should be tested. If you do not want to tell your partners yourself, the outreach workers will contact them, according to the privacy guidelines of the [health authority].

# RESEARCH-RELATED INJURY

[Sites to specify institutional policy:] It is unlikely that you will be injured because of your study participation. If you are injured, the [institution] will give you immediate necessary treatment for your injuries. You [will/will not] have to pay for this treatment. You will be told where you can get further treatment for your injuries. There is no program to pay money or give other forms of compensation for such injuries either through this institution or the US NIH. You do not give up any legal rights by signing this consent form.

## PROBLEMS OR QUESTIONS

If you ever have any questions about the study, or if you have a research-related injury, you should contact [insert name of the investigator or other study staff] at [insert telephone number and/or physical address].

If you have questions about your rights as a research participant, you should contact [insert name or title of person on the IRB or other organization appropriate for the site] at [insert physical address and telephone number].

# **SIGNATURE PAGE**

Enhancing Recruitment, Linkage to Care and Treatment for HIV-Infected Men Who Have Sex with Men (MSM) in the United States

# **HPTN 078**


# ENROLLMENT INFORMED CONSENT FORM

If you have read this consent form, or had it read and explained to you, and you understand the information, and you voluntarily agree to join the study, please sign your name or make your mark below.

| Participant Name (print) | Participant Signature and Date |
|---|---|
| Study Staff Conducting Consent Discussion (print) | Study Staff Signature and Date |
| Witness Name (print) (As appropriate) | Witness Signature and Date |

# SIGNATURE PAGE FOR PARTICIPANTS BELOW THE LEGAL AGE TO PROVIDE INDEPENDENT INFORMED CONSENT

Enhancing Recruitment, Linkage to Care and Treatment for HIV-Infected Men Who Have Sex with Men (MSM) in the United States

# **HPTN 078**


# ENROLLMENT INFORMED CONSENT FORM

| Participant Assent | |
|---|---|
| | or had it read and explained to you, and you understand the gree to join the study, please sign your name or make your |
| Participant Name (print) | Participant Signature and Date |
| Parent/Legal Guardian Consent | |
| | or had it read and explained to you, and you understand the gree for your child to join the study, please sign your name o |
| Parent/Guardian Name (print) | Parent/Guardian Signature and Date |
| Study Staff Conducting Consent Discussion (print) | Study Staff Signature and Date |
| Witness Name (print) | Witness Signature and Date |

(As appropriate)

# **Enhancing Recruitment, Linkage to Care and Treatment for HIV-Infected Men Who Have Sex with Men (MSM) in the United States**

## **HPTN 078**


# SAMPLE STORAGE AND FUTURE USE CONSENT FORM

**Sponsored by:** Division of AIDS (DAIDS), United States (US) National Institute of Allergy and Infectious Diseases (NIAID), US National Institute of Mental Health (NIMH), US National Institute on Drug Abuse (NIDA) and US National Institutes of Health (NIH).

PRINCIPAL INVESTIGATOR: [Insert Name]

**PHONE:** [Insert Number]

#### POSSIBLE FUTURE TESTS

If you give permission, some of the plasma (a part of the blood) collected from you will be kept after the study ends for possible testing related to HIV and hepatitis C virus and to better understand laboratory tests related to this study. If you do not agree to have your left over plasma stored you can still be in this study. If you agree to store your plasma but change your mind later, you can contact study staff. We will then destroy your samples. If you agree, your left over plasma will be stored for at least three years after the study ends. Any future use, not related to HIV or hepatitis C virus, needs to be reviewed and approved by the NIH and local authorities. Your left over samples will not be sold or used for commercial reasons.

# **SIGNATURE PAGE**

# Enhancing Recruitment, Linkage to Care and Treatment for HIV-Infected Men Who Have Sex with Men (MSM) in the United States

# **HPTN 078**


# SAMPLE STORAGE AND FUTURE USE CONSENT FORM

If you have read this consent form, or had it read and explained to you, and you understand the information, and you voluntarily agreed to join the study, please sign your name or make your

My initials indicate that some of the plasma collected from me may be stored for future testing after study-related testing has been completed.

\_\_\_\_\_ I do not agree to allow left over plasma samples to be saved for long-term storage or future testing after study-related testing has been completed.

Participant Name (print) Participant Signature Date

Study Staff Conducting Study Staff Signature Date

Consent Discussion (print)

# SIGNATURE PAGE FOR PARTICIPANTS BELOW THE LEGAL AGE TO PROVIDE INDEPENDENT INFORMED CONSENT

Enhancing Recruitment, Linkage to Care and Treatment for HIV-Infected Men Who Have Sex with Men (MSM) in the United States

# **HPTN 078**


# SAMPLE STORAGE AND FUTURE USE CONSENT FORM

| Participant Assent | |
|---|---|
| 2 | r had it read and explained to you, and you understand the eed to join the study, please sign your name or make your |
| My initials indicate that some testing after study-related testing has | e of the plasma collected from me may be stored for future been completed. |
| I do not agree to allow left ov future testing after study-related testing | ver plasma samples to be saved for long-term storage or ng has been completed. |
| Participant Name (print) | Participant Signature and Date |
| Parent/Legal Guardian Consent | |
| 2 | had it read and explained to you, and you understand the sed for your child to join the study, please sign your name or |
| Parent/Guardian Name (print) | Parent/Guardian Signature and Date |
| Study Staff Conducting Consent Discussion (print) | Study Staff Signature and Date |
| Witness Name (print) | Witness Signature and Date |

(As appropriate)

# Enhancing Recruitment, Linkage to Care and Treatment for HIV-Infected Men Who Have Sex with Men (MSM) in the United States

## **HPTN 078**


## EXIT INTERVIEW FOR CASE MANAGERS CONSENT FORM

**Sponsored by:** Division of AIDS (DAIDS), United States (US) National Institute of Allergy and Infectious Diseases (NIAID), US National Institute of Mental Health (NIMH), US National Institute on Drug Abuse (NIDA) and US National Institutes of Health (NIH).

PRINCIPAL INVESTIGATOR: [Insert Name]

**PHONE:** [Insert Number]

#### INTRODUCTION

You are being asked to take part in a research study that is designed to find out if support from a case manager can help HIV-infected people receive consistent HIV care and routinely take their HIV medication. Joining this study is voluntary. You may refuse to join, or you may withdraw your consent to be in the study, for any reason. As part of the study, you are being asked to take part in an exit interview.

Before you decide whether to join the study, we would like to explain the purpose of the study, the risks and benefits to you, and what is expected of you.

# YOUR PARTICIPATION IS VOLUNTARY

This consent form gives information about the study you are being invited to join. Once you understand the study, and if you agree to take part, you will be asked to sign your name or make your mark on this form. You will be offered a copy of this form to keep.

Before you learn about the study, it is important that you know the following:

- Your participation is voluntary. You do not have to take part in the exit interview.
- You may decide to leave the exit interview at any time.
- If you decide not to take part in the exit interview, you can still join another study at a later time if there is one available and you qualify.
- If you decide not to take part in the exit interview, or decide to stop participating at any time, there will be no penalty or loss of normal benefits provided to you at our clinic.

## PURPOSE OF THE STUDY

The purpose of this study is to find out if support from a case manager can help HIV-infected people receive consistent HIV care and routinely take their HIV medication.

# STUDY PROCEDURES

If you decide to join the study, you will be asked to participate in an exit interview at the end of the study. This interview may include both a questionnaire to complete as well as a semi-structured interview (by talking to the interviewee). Both the questionnaire and the interview will ask you about your experience and opinions in administering the CM intervention in this study.

# RISKS AND/OR DISCOMFORTS

# **Sensitive Questions**

It is possible that the questions about your experience in administering the CM intervention may make you feel uneasy. However, you do not have to answer any question that you do not want to and you can stop answering the questions at any time.

# **BENEFITS**

You may not receive any direct benefit from being in this study. The information gathered during this study may help prevent HIV in the MSM community.

## **NEW INFORMATION**

You will be told about any new information learned during this study that might affect your willingness to take part in the study. You will also be told when the results of the study may be available, and how to learn about them.

#### WHY YOU MAY BE WITHDRAWN FROM THE STUDY WITHOUT YOUR CONSENT

You may be withdrawn from the study without your consent if any of the following occur:

- You are unable or unwilling to follow the study procedures or instructions.
- The study is stopped or canceled.
- The study staff feels that staying in the study would be harmful to you.
- Other reasons, as decided by the study staff.

#### ALTERNATIVES TO PARTICIPATION

You may choose not to participate in the study. [Sites to include/amend the following if applicable: There may be other studies going on here or in the community that you may be eligible for. If you wish, we will tell you about other studies that we know about.]

## **COSTS TO YOU**

There will be no cost to you for this interview.

#### REIMBURSEMENT

You will receive [site to add amount] for your time and effort for this interview. [Sites to insert information about local reimbursement for the study.]

# **CONFIDENTIALITY**

All the information you give us as part of this study will be kept private. You will get a unique study identification number that will be used instead of your name on your documents. Only the study staff will be able to see records that identify you by name. This information will not be shared with others. All records will be stored in locked files at the study clinic. Your name will never be used in any publication or presentation about the study.

Your records may be reviewed by the sponsor of the study, the US National Institutes of Health (NIH) and their representatives, other government and regulatory authorities, [insert name of site] IRB/EC, study staff, study monitors and [insert applicable local regulatory authorities].

In addition to the efforts made by the study staff to help keep your personal information confidential, we have obtained a Certificate of Confidentiality from the U.S. Federal Government. This Certificate protects researchers from being forced to tell people who are not connected with this study, such as the court system, about your participation. The Certificate of Confidentiality does not prevent you from releasing information about yourself and your participation in the study. The Certificate cannot be used to resist a demand for information from personnel of the US Government that is used for auditing or evaluation of federally funded projects or for information that must be disclosed in order to meet the requirements of the US FDA. Even with the Certificate of Confidentiality, if the study staff learns of possible child abuse and/or neglect or a risk of harm to you or others, we will tell the proper authorities.

A description of this study will be available on <u>www.ClinicalTrials.gov</u>. This web site will not include information that can identify you. At most, the web site will include a summary of the results. You can search this web site at any time.

# RESEARCH-RELATED INJURY

[Sites to specify institutional policy:] It is unlikely that you will be injured as a result of study participation. If you are injured, the [institution] will give you immediate necessary treatment for your injuries. You [will/will not] have to pay for this treatment. You will be told where you can get additional treatment for your injuries. There is no program to pay money or give other forms of compensation for such injuries either through this institution or the US NIH. You do not give up any legal rights by signing this consent form.

# PROBLEMS OR QUESTIONS

If you ever have any questions about the study, or if you have a research-related injury, you should contact [insert name of the investigator or other study staff] at [insert telephone number and/or physical address].

If you have questions about your rights as a research participant, you should contact [insert name or title of person on the IRB or other organization appropriate for the site] at [insert physical address and telephone number].

# **SIGNATURE PAGE**

Enhancing Recruitment, Linkage to Care and Treatment for HIV-Infected Men Who Have Sex with Men (MSM) in the United States

## **HPTN 078**


# EXIT INTERVIEW FOR CASE MANAGERS CONSENT FORM

If you have read this consent form, or had it read and explained to you, and you understand the information, and you voluntarily agree to participate in the exit interview, please sign your name or make your mark below.

| Participant Name (print) | Participant Signature and Date |
|---|---|
| Study Staff Conducting Consent Discussion (print) | Study Staff Signature and Date |
| Witness Name (print) (As appropriate) | Witness Signature and Date |

| APPENDIX IV: TAILORED CASE MANAGEMENT INTERVENTION COMPONENTS<br>IN AT RISK US POPULATIONS(2005 – 2015) |
|---|

| HPTN 078<br>CM<br>Intervention<br>Component | First Author;<br>Year;<br>Location(s) | Design;<br>Sample Size | Study Focus /<br>Intervention<br>Component(s) | Evidence of Effect | Cascade<br>Component |
|---|---|---|---|---|---|
| | Yehia; 2015;<br>Philadelphia,<br>PA <sup>51</sup> | Cross Sectional; Descriptive; 1359 newly HIV diagnosed adults Qualitative; 30 | Testing location Self determination | <ul> <li>Testing/diagnosis locations without colocated outpatient care are associated with delayed linkage to care</li> <li>Counseling and testing centers, correctional centers, and inpatient settings are found to delay linkage to care in comparison to medical clinics</li> <li>Medical clinics integrate testing and medical services, facilitating linkage to care (decreased wait times, increased familiarity with facilities, supportive ancillary services)</li> <li>Autonomy is lost at diagnosis due to</li> </ul> | - Linkage to care - Engagement in care - Linkage to care |
| My Life | Chapel Hill, NC <sup>49</sup> | HIV-positive<br>women of<br>color | theory in HIV | stigma, feelings of helplessness, and lack of competency. Autonomy/self-motivation and competency should be regained to facilitate engagement in care - Welcoming environment at initial clinical encounter would influence support and self-motivation to return for following visits - Increasing health-related knowledge and healthcare navigation facilitates feelings of competency - Retention in care is influenced by strong relationships between providers and patients, but long-term engagement is most influenced by developing autonomy and self-management | - Retention in care - Self- management - Durability |

July 3, 2017  HPTN 078, Final Version 2.0

| HPTN 078<br>CM<br>Intervention<br>Component | First Author;<br>Year;<br>Location(s) | Design;<br>Sample Size | Study Focus /<br>Intervention<br>Component(s) | Evidence of Effect | Cascade<br>Component |
|---|---|---|---|---|---|
| | Hightow; 2011;<br>Chapel Hill, NC <sup>48</sup> | Pre-post test;<br>81 HIV-<br>positive MSM<br>of color | Linkage to care program including: - Social marketing - Intense outreach - Medical/social support | <ul> <li>76% viral suppression at 12 months</li> <li>Odds of 1 clinic visit in 4 months post-intervention versus pre-intervention group (OR = 2.58; 95% CI 1.34 – 4.98)</li> <li>Likelihood of clinic visit attendance decreased over time for both pre- and post-intervention groups, yet for the intervention group retention was significantly greater</li> </ul> | <ul> <li>Linkage to care</li> <li>Retention in care</li> <li>Viral<br/>suppression</li> <li>Durability</li> </ul> |
| My Life<br>(cont) | Rajabiun; 2007;<br>6 cities from<br>northwest,<br>midwest,<br>midatlantic and<br>northeast regions | Qualitative;<br>purposive<br>sampling; 76<br>HIV-positive<br>adults;<br>26% MSM | Interviews to understand participants' experiences with engagement and retention | <ul> <li>Participants cycle in and out of care and this process is facilitated or obstructed by the relationship of the patient with the provider</li> <li>Partnership, validation, trust, respect, and emotional intelligence were notable characteristics of providers who influenced patients to engage and remain in care</li> <li>When patients felt that their provider was patronizing or that they encountered stigma, they were less likely to remain in care</li> <li>Engagement depends upon: <ul> <li>Acceptance level of diagnosis</li> <li>Ability to cope with substance abuse, mental illness and stigma</li> <li>Healthcare provider relationships</li> <li>External support systems</li> <li>Ability to overcome practice barriers to care</li> </ul> </li> </ul> | <ul> <li>Linkage to care</li> <li>Retention in care</li> <li>Engagement in care</li> <li>Inter-personal relationship building</li> </ul> |

July 3, 2017  HPTN 078, Final Version 2.0

| HPTN 078<br>CM<br>Intervention<br>Component | First Author;<br>Year;<br>Location(s) | Design;<br>Sample Size | Study Focus /<br>Intervention<br>Component(s) | Evidence of Effect | Cascade<br>Component |
|---|---|---|---|---|---|
| My Choices | Craw; 2010;<br>Anniston, AL<br>Atlanta, GA<br>Baltimore, MD<br>Baton Rouge, LA<br>Chicago, IL<br>Columbia, SC<br>Jacksonville, FL<br>Kansas City, MO<br>Miami, FL<br>Richmond, VA <sup>53</sup> | ARTAS II<br>demonstration<br>project;<br>626 HIV-<br>positive adults | Strengths-Based Linkage Case Management; Identify barriers and solutions to overcome challenges to engagement in care | <ul> <li>79% (497 of 626) of participants visited an HIV clinician at least once within the first 6 months</li> <li>Number of case management sessions (2-5 sessions) was associated with greater linkage (OR = 2.95, 95% CI 1.88 – 4.62)</li> <li>Mean time spent per client was 7.2; median 5.8 hours</li> <li>Biggest barriers to engagement by patient self report were 1) feeling well; 2) lack of transport; 3) not ready to start HIV medications; 4) no insurance; 5) took too long to get an appointment</li> <li>Durability of project was limited due to lack of funding</li> <li>Those sites that continued the linkage program after funding ended had long-standing relationships with local health departments and a steady influx of HIV patients</li> </ul> | - Linkage to care - Engagement in care |
| | Christopoulos;<br>2013;<br>San Francisco,<br>CA <sup>52</sup> | Qualitative; 34<br>HIV-positive<br>adults;<br>55% MSM | Qualitative<br>interviews around<br>engagement and<br>linkage in newly<br>diagnosed | <ul> <li>Linkage to care experience lays groundwork for subsequent retention in care</li> <li>All patients reported have to learn and manage the "administrative" aspects of care in order to stay engaged in care</li> <li>Patient priorities change over time, often shifting from medical/physical concerns to psychological/social concerns – interventions must</li> </ul> | <ul> <li>Linkage to care</li> <li>Engagement in care</li> <li>Retention in care</li> </ul> |


July 3, 2017


| HPTN 078<br>CM<br>Intervention<br>Component | First Author;<br>Year;<br>Location(s) | Design;<br>Sample Size | Study Focus /<br>Intervention<br>Component(s) | Evidence of Effect | Cascade<br>Component |
|---|---|---|---|---|---|
| | , | Prospective cohort; 437 HIV-positive adults Descriptive, observational; 5631 HIV-positive adults | | accommodate this shift in order to continue to engage patients in care Relationship building noted in 86% Navigation services were used in 74% Participants who had improved engagement with their provider had "41% greater odds of undetectable viral load" and 32% "greater odds of reporting the optimal number of HIV visits at 12 months" 56.7% received care at MCM-funded facilities of which 76.2% (vs. 59.9% in non-MCM funded facilities) were retained in care, and 70.6% (vs. 75.7%) achieved viral suppression. Those receiving care in MCM-funded facilities more likely to be retained in care (aOR 4.13; 95%CI: 1.93-8.85) and as likely (aOR 1.06; 95%CI: 0.68-1.62) to be virally suppressed. Among 789 newly diagnosed persons, those diagnosed in MCM-funded facilities were not more likely to be linked to care within 3 months (aOR 0.50; 95%CI: 0.21-1.18). | - Engagement in care - Retention in care - Viral suppression - Durability - Linkage to care - Engagement in care - Retention in care - Viral suppression - |

July 3, 2017  HPTN 078, Final Version 2.0

| HPTN 078<br>CM<br>Intervention<br>Component | First Author;<br>Year;<br>Location(s) | Design;<br>Sample Size | Study Focus /<br>Intervention<br>Component(s) | Evidence of Effect | Cascade<br>Component |
|---|---|---|---|---|---|
| | Naar-King; 2009;<br>Detroit, MI <sup>60</sup> | Pilot<br>randomized<br>trial; 87 HIV-<br>positive youth<br>(16 – 29) | Motivational interviewing by peer versus professional | <ul> <li>Peer and professional interviewers had similar motivational interviewing scores</li> <li>Established initial effect size for peerbased MI programs</li> <li>Both groups improved the regularity of primary care HIV appointments</li> <li>Peer outreach is a cost-effective and durable program</li> </ul> | <ul><li>Retention in care</li><li>Durability</li></ul> |
| My Care<br>(Step 2) | Hayley; 2014;<br>New York City,<br>NY<br>Newark, NJ<br>Washington DC<br>Baltimore, MD<br>Durham, NC<br>Atlanta, GA <sup>58</sup> | Prospective,<br>observational<br>cohort;<br>2099 HIV-<br>negative<br>women at risk<br>of HIV<br>acquisition | Interpersonal relationship building; community engagement; reduction of external barriers; staff capacity building participant tracing | <ul> <li>Participant visit completion was 93% at 6 months</li> <li>Participant visit completion was 94% at 12 months</li> <li>Housing instability was a significant predictor of missed visits</li> </ul> | <ul> <li>Engagement in care</li> <li>Retention in care</li> <li>Inter-personal relationship building</li> <li>Durability</li> </ul> |
| | Remien; 2005;<br>New York City,<br>NY <sup>62</sup> | Randomized controlled trial; 215 sero-discordant couples with suboptimal adherence | 4 session, couple focused adherence to medication intervention | <ul> <li>Higher medication adherence post-intervention in proportion of prescribed doses taken (76% versus 60%)</li> <li>Greater likelihood of high levels of adherence compared to controls</li> <li>Effects diminish with time</li> <li>No significance difference identified between increased adherence and viral suppression</li> <li>Involvement of relationship partner in treatment decisions and adherence is durable, cost-effective and improves adherence and treatment support</li> </ul> | <ul> <li>Engagement in care</li> <li>Adherence</li> <li>Retention in care</li> <li>Durability</li> </ul> |

July 3, 2017  HPTN 078, Final Version 2.0

| HPTN 078<br>CM<br>Intervention<br>Component | First Author;<br>Year;<br>Location(s) | Design;<br>Sample Size | Study Focus /<br>Intervention<br>Component(s) | Evidence of Effect | Cascade<br>Component |
|---|---|---|---|---|---|
| | Simoni; 2006;<br>Multisite <sup>32</sup> | Meta analysis;<br>19 studies;<br>1839 HIV-<br>positive<br>participants;<br>53% MSM<br>(median across<br>all studies) | Randomized<br>behavioral<br>interventions<br>in adults | <ul> <li>Behavioral interventions (e.g. education, cognitive behavioral therapy, motivational interviewing, group therapy, cue dosing) increased 95% adherence (OR = 1.50; 95% CI 1.16 – 1. n = 1633), but did not meet statistical significance for undetectable viral load (OR = 1.25; 95% CI 0.99 – 1.59; n = 1247)</li> <li>In the sub-analysis that evaluated studies with 50% of greater MSM, the results for viral load were OR = 1.83; 95% CI 0.50 – 6.67)</li> </ul> | <ul><li>Adherence (self-report)</li><li>Viral suppression</li></ul> |
| My Care<br>(Step 2)<br>(cont) | Nelsen; 2013;<br>Houston, TX <sup>61</sup> | Cross-<br>sectional<br>survey; 244<br>HIV-positive<br>adults | Patient intention<br>to adhere to HIV<br>treatment | - Intention to adhere (measured by the 13-item Intention to Adhere to HIV Treatment Scale) was the only "patient-centered" outcome that predicated adherence (OR 2.2; 95% CI 1.1 – 4.3) | - Adherence |
| | Holtzman; 2015;<br>Philadelphia,<br>PA <sup>59</sup> | Qualitative<br>semi-<br>structured<br>interviews; 51<br>HIV-positive<br>adults | Andersen's<br>Behavioral Model | <ul> <li>Low retention and adherence was predicted by stigma, mental illness, substance abuse, low social support, poor reminder strategies, housing, insurance, symptoms, competing life activities, colocation of services, and provider factors</li> <li>Barriers specific to retention included transportation, clinic experiences, and appointment scheduling</li> <li>Barriers specific to adherence included medication characteristics, pharmacy services, health literacy, and health benefits</li> </ul> | - Retention in care - Adherence |

July 3, 2017  HPTN 078, Final Version 2.0

| HPTN 078<br>CM<br>Intervention<br>Component | First Author;<br>Year;<br>Location(s) | Design;<br>Sample Size | Study Focus /<br>Intervention<br>Component(s) | Evidence of Effect | Cascade<br>Component |
|---|---|---|---|---|---|
| | Lewis; 2013;<br>Midwest HIV<br>Clinic <sup>38</sup> | Pre- experimental proof of concept study; 52 HIV- positive MSM | Pre-post test design; Tailored text messaging intervention | <ul> <li>Positive receptivity to text messages, both in content and frequency</li> <li>Overall, participants had an improvement in viral load control (&lt;75) and CD4 count</li> <li>Decrease in number of missed medication days</li> <li>Message fatigue was common but could be addressed through customizing and varying the messages delivered to make the intervention more durable</li> </ul> | <ul> <li>Adherence</li> <li>Self- management</li> <li>Inter-personal relationship building</li> <li>Viral suppression</li> <li>Durability</li> </ul> |
| My Health | Schnall; 2015;<br>New York City <sup>57</sup> | Focus Groups;<br>50 PLWH | technology | <ul> <li>Participants suggested several tools for meeting their healthcare needs, including: reminders/alerts, lab results tracking, and notes on health status.</li> <li>mHealth technology can function as a social actor by providing chat boxes/forums, testimonials of lived experiences, and personal outreach.</li> <li>Examples of media that can be used as a persuasive technology include games/virtual rewards, coding of health tasks, and simulations on how to interact and connect with others</li> </ul> | - Adherence - Self management |

July 3, 2017  HPTN 078, Final Version 2.0

| HPTN 078<br>CM<br>Intervention<br>Component | First Author;<br>Year;<br>Location(s) | Design;<br>Sample Size | Study Focus /<br>Intervention<br>Component(s) | Evidence of Effect | Cascade<br>Component |
|---|---|---|---|---|---|
| My Health (cont) | Hightow; 2011; Chapel Hill, NC; Bronx, NY; Chicago, IL; Detroit, MI; Houston, TX; Los Angeles, CA; Oakland, CA; Rochester, NY <sup>55</sup> Gilman; 2012; five sites from the Northeast, Midwest, and the South <sup>54</sup> | Site visits; seven linkage programs in five sites | National HIV/AIDS Bureau program: Outreach, linkage, entry, and retention analysis Hospital-based, integrated linkage to care programs | <ul> <li>Earlier linkage to care was significantly associated with the person who made the diagnosis also making the initial referral to care</li> <li>Clinic appointment reminders, case finding for patients who had missed appointments, transportation assistance as well as dedicated providers were all factors that contributed to the high retention rate of 83% of participants at one year</li> <li>Dedicated providers contributed to the sustainability of the program</li> <li>Successful linkage programs are low cost, intensive, time limited, flexible, and unique</li> <li>Successful programs directly employed linkage workers, actively referred newly diagnosed patients to medical care, employed person-centered case management, and were culturally and linguistically in concordance with populations served</li> <li>Successful implementation of linkage programs requires coordination and integration of services among testing and treatment sites, sustaining funding sources, and ensuring commitment from program stakeholders and testing staff</li> </ul> | - Linkage to care - Durability - Linkage to care - Durability |


July 3, 2017


| HPTN 078 CM Intervention Component | First Author;<br>Year;<br>Location(s) | Design;<br>Sample Size | Study Focus /<br>Intervention<br>Component(s) | Evidence of Effect Cascade Component |
|---|---|---|---|---|
| My Health<br>(cont) | Maulsby; 2015;<br>Chicago, IL; New<br>York City, NY;<br>Louisiana <sup>56</sup> | Descriptive;<br>2,615 HIV<br>positive adults | Positive Charge<br>HIV linkage and<br>re-engagement in<br>care program | <ul> <li>Through methods such as peer health navigation, peer-led group-based education, case management, and case finding 88% of participants were linked to care, 69% were retained in care and 46% were virally suppressed at follow-up</li> <li>90% of MSM in one site were engaged in care following enrollment</li> <li>Sustainable programs targeting underserved populations are achievable</li> </ul> |


July 3, 2017
